

# Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

| Document Number: | c39712001-02 |
|---|---|
| BI Study Number: | 1245-0228 |
| BI Investigational<br>Product(s) | Jardiance® (empagliflozin) |
| Title: | Comparative cardiovascular and renal effectiveness and safety of Empagliflozin and other SGLT2i in patients with type 2 diabetes (T2D), with and without baseline kidney disease in the United States: Statistical an Epidemiological Analysis Plan |
| Brief lay title: | Evaluating comparative effectiveness of empagliflozin in patients with type 2 diabetes with and without chronic kidney disease |
| SEAP version identifier: | 2.0 |
| Date of last version of SEAP: | 8 July 2022 |
| Date of current version of SEAP: | 28 July 2023 |
| NIS Statistician [SEAP author] | |
| NIS [SEAP reviewer] | |
| NIS Data [SEAP reviewer] | |


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

**BI Study Number 1245-0228** 

c39712001-02



Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 1. TABLE OF CONTENTS

| ΤI | TLE PAGE | | 1 |
|---|---|---|---|
| 1. | TABLE O | F CONTENTS | 3 |
| 2. | LIST ABE | BREVIATIONS | 5 |
| 3. | RESPONS | SIBLE PARTIES | 7 |
| 4. | PURPOSE | E AND SCOPE | 8 |
| 5. | AMENDM | MENTS AND UPDATES | 9 |
| 6. | RESEARC | CH QUESTION AND OBJECTIVE | 10 |
| 7. | RESEARC | CH METHODS | 11 |
| | 7.1 | STUDY DESIGN | 11 |
| | 7.2 | SETTING | 11 |
| | 7.3 | STUDY PERIOD | 11 |
| | 7.4 | STUDY POPULATION | 11 |
| | 7.4.1 | Inclusion and exclusion criteria. | 12 |
| | 7.4.2 | Preliminary patient counts | 13 |
| | 7.5 | STUDY VISITS | 14 |
| | 7.5.1 | Baseline period (lookback period) | 14 |
| 8. | VARIABI | LES | 15 |
| | 8.1 | Exposures | 15 |
| | 8.1.1 | Study medications | 16 |
| | 8.1.2 | Operational definitions on how to identify each of the index medication | |
| | cohorts | | |
| | 8.1.3 | Definition of censored follow-up end | |
| | 8.2 | Outcomes | |
| | 8.2.1 | Primary outcomes | |
| | 8.2.2 | Secondary outcomes. | 20 |
| | 8.3 | Covariates | 22 |
| 9. | | URCES | |
| 9.<br>10 | | MANAGEMENT AND SOFTWARE/TOOLS | |
| 10 | 10.1 | Software/Tools | |
| | 10.1 | Handling of Missing Values. | |
| | 10.4 | TIMIMITIE OF INTEGRAL A MINOR AND THE PROPERTY OF THE PROPERTY | |

| 0 | r Ingelheim<br>and Epidemiological Analysis Plan (SEAP) for Non-Inter | Page 4 of 40<br>ventional Study |
|---|---|---|
| | Number 1245-0228 | c39712001-02 |
| Proprietary | confidential information © 2023 Boehringer Ingelheim International GmbH or one or more | e of its affiliated companies |
| 10.3 | Handling of Inconsistencies in Data and Outliers | 33 |
| 11. DA | TA ANALYSIS | 34 |
| 11.1 | Phased Approach | 34 |
| 11.2 | Propensity score models and overlap weighting | 34 |
| 11.3 | Descriptive analyses | 35 |
| 11.4 | Comparative effectiveness analyses | 35 |
| 11.4.1 | Empagliflozin vs. DPP4i | 35 |
| 11.4.2 | SGLT2i vs. GLP1RA | 36 |
| 11.6 | Safety Analysis | 38 |
| 12. QU | ALITY CONTROL | 39 |
| 13. REI | FERENCES | 40 |
| 13.1 | PUBLISHED REFERENCES | 40 |
| 13.2 | UNPUBLISHED REFERENCES | 40 |
| 14. AN | NEXES | 41 |
| ANNEX 1. | LIST OF STANDALONE DOCUMENTS | 41 |
| ANNEX 2. | PROPOSED TABLES AND FIGURES | 42 |
| ANNEX 3. | REVIEWERS AND APPROVAL SIGNATURES | 69 |
| ANNEX 4 | CODFLIST | 70 |


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

(NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. LIST ABBREVIATIONS

ACD All-Cause Death

ADR Adverse Drug Reaction

AE Adverse Event

AESI Adverse Event of Special interest

AKI Acute Kidney Injury

ASMD Absolute Standardized Mean Difference

AT As-Treated

AV Ambulatory Visit

BI Boehringer Ingelheim
CA Competent Authority

CCDS Company Core Data Sheet

CDM Common Data Model
CI Confidence Interval

CML Local Clinical Monitor

CRA Clinical Research Associate

CRF Case Report Form

CTCAE Common Terminology Criteria for Adverse Events

CTP Clinical Trial Protocol

CV Cardiovascular

DKD Diabetic Kidney Disease

DMRP Data Management and Review Plan

DPP4i Dipeptidyl Peptidate-4 inhibitor

eCRF Electronic Case Report Form

ED Emergency Department
EHR Electronic Health Record

ENCePP European Network of Centres for Pharmacoepidemiology and

Pharmacovigilance

ESRD/ESKD End Stage Renal (Kidney) Disease

FDA Food and Drug Administration

GCP Good Clinical Practice


## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

(NIS)

## **BI Study Number 1245-0228**

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

GEP Good Epidemiological Practice

GLP1RA Glucagon-like Peptide-1 Receptor Agonists

GPP Good Pharmacoepidemiology Practice

GVP Good Pharmacovigilance Practices

HF Heart Failure
HR Hazard Ratio

IB Investigator's Brochure

IEC Independent Ethics Committee

IQR Interquartile Range

IRB Institutional Review Board

ITT Intent-to-treat

MAH Marketing Authorization Holder

MedDRA Medical Dictionary for Regulatory Activities

NIS Non-Interventional Study

PASS Post-Authorization Safety Study

PCORnet Patient Centered Outcomes Research Network

PS Propensity Score
QC Quality Control

SAE Serious Adverse Event

SEAP Statistical and Epidemiological Analysis Plan SGLT2i Sodium glucose co-transporter-2 inhibitors

SOP Standard Operating Procedure

SSDC Study Specific Data Characterization

T1D Type 1 Diabetes Mellitus
T2D Type 2 Diabetes Mellitus

TH Telehealth Visit

UTI Urinary Tract Infection


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. RESPONSIBLE PARTIES

Non-interventional study (NIS) Statistician (statistical epidemiological analysis plan [SEAP] author):

Other supporting parties:

| Name, degree(s) | Title | Affiliation | Address |
|---|---|---|---|
| | Global<br>Epidemiologist | Boehringer<br>Ingelheim<br>International GmbH | |
| | Global RWE<br>Analytics Center<br>of Excellence | Boehringer<br>Ingelheim<br>International GmbH | |
| | Statistical<br>Research Scientist | | |
| | Informaticist | | |
| | Investigator | | |
| | Co-investigator | | |

- BI NIS [SEAP reviewer] (in all cases): Global Epidemiology
- NIS Data [SEAP reviewer] (in all cases):
- RWE CoE [SEAP reviewer] (for all globally initiated studies and for local studies) involving BI products and Global NIS not involving BI products: World Evidence CoE
- TSTAT (for NISnd only): Not Applicable
- TM Epi [SEAP reviewer] (When BI NIS lead is not TM Epi; in all cases): Not Applicable

BI Study Number 1245-0228

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c39712001-02

## 4. PURPOSE AND SCOPE

SEAP reviewers are expected to be familiar with the NIS protocol entitled "Comparative cardiovascular and renal effectiveness and safety of Empagliflozin and other SGLT2i in patients with type 2 diabetes (T2D), with and without baseline kidney disease in the United States", version 1.0 dated 10 June 2022 unless otherwise stated.

The SEAP addresses the details of the implementation of this study. In the SEAP, you can find operational definitions on how to identify each of the index medication cohorts, detailed data analysis plan such as the propensity score weighting, and main analysis plan. In addition, the study codelists are captured in the accompanying document entitled 1245.0228 Empa DKD Codelist Master with Sources 15June2023.xlsx.


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 5. AMENDMENTS AND UPDATES

| Amendment<br>Number | Date | Section of<br>the study<br>protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 1 | 26 May 2023 | 5.0<br>6.0<br>7.0 | Removal of analyses involving comparison of empagliflozin vs GLP1RA. | Phase 1 analyses indicated differences in treatment exposure between patients prescribed empagliflozin compared to those prescribed GLP1RAs (i.e., greater proportion of patients prescribed 4+ prescriptions observed for GLP1RA over follow up) |
| 2 | 26 May 2023 | 7.0 | Added study outcome | The composite outcome of MI + stroke+all-cause death+ cardiovascular revascularization was previously in the protocol but the composite MI+stroke +all-cause death was added |
| 3 | 26 May 2023 | 10.5 | Addition of acute<br>HHF codes as a<br>sensitivity analysis | The initial broader codelist for HHF will be performed but a sensitivity analysis only including HHF that indicate acute HF will be examined. |


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 6. RESEARCH QUESTION AND OBJECTIVE

## **Primary Objective:**

- To determine the cardiovascular and renal effectiveness and safety of empagliflozin compared to dipeptidyl peptidase 4 inhibitor (DPP4i) in patients with type 2 diabetes (T2D) in the
  - o Overall cohort,
  - o Patients with established kidney disease (DKD cohort), and
  - O Patients without established kidney disease (non-DKD cohort).

## Secondary Objective:

• To determine the cardiovascular and renal effectiveness and safety of any sodiumglucose co-transporter-2 inhibitor (SGLT2i) compared to glucagon-like peptide-1 receptor agonist (GLP1RA).


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. RESEARCH METHODS

#### 7.1 STUDY DESIGN

This will be a non-interventional study (NIS) using existing data from up to 20 US healthcare systems that have mapped their electronic health record (EHR) data to the PCORnet Common Data Model (CDM).<sup>1</sup>

The study uses a "new users" design and compares patients initiating empagliflozin or other SGLT2i to initiators of DPP4i. Additionally, the feasibility of also including GLP1RA as a comparison group will be examined. The comparator group(s) have the same indication as that of the empagliflozin or SGLT2i group and comparator medications were potentially prescribed to patients with T2D with similar characteristics; that is, similar T2D severity and underlying diabetes-related comorbidities after propensity score overlap weighting will be performed between new users of empagliflozin compared to DDP4i and SGLT2i compared to GLP1RA comparison groups.

## 7.2 SETTING

The data sources included in the study will be participating health systems from PCORnet in the United States (US) and Datavant. For further details on this data sources, please see **Section 9** in the study protocol.

## 7.3 STUDY PERIOD

The study period will be from 1 January 2014 through 31 December 2021, which includes data after the start of the COVID-19 pandemic. There will be an assessment of COVID-era data for quality purposes and a sensitivity analysis excluding data from March 2020 to the end of study period will be performed.

#### 7.4 STUDY POPULATION

The study population will include adults with T2D that are new users of empagliflozin compared to new users of a DPP4i or new users of SGLT2i compared to new users of GLP1RA. New users will be defined as those having a prescription of a study medication during the study period and who have not received a prescription of either of the study medications during the 12 months before the index date (specific to each comparison). The date of the first prescription of a study medication of interest within the study period which meet all the inclusion criteria will be the index date.

Codes to select study populations are provided in accompanying document 1245.0228 Empa DKD Codelist Master with Sources 15June2023.xlsx.

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.4.1 Inclusion and exclusion criteria

The analyses will include adults (≥18 years) with T2D with or without kidney disease in the US. To study real-world treatment patterns, the study population will include a broad spectrum of patients initiating empagliflozin, any SGLT2i, any DPP4i, or any GLP1RA. The following inclusion and exclusion criteria will be used for each two-arm comparison:

Included patients will be required to meet *all* the following criteria:

- Patients  $\geq$ 18 years old,
- Having a diagnosis of T2D within 12 months prior to the index date (defined as the date of initiation of empagliflozin or any SGLT2i, any GLP1RA, or any DPP4i based on the cohort evaluated) based on ICD-9 and ICD-10 codes,
- Record of 1+ prescription for empagliflozin, any SGLT2i, any DPP4 inhibitor, or any GLP1RA use between 1 January 2015 and 31 December 2020, and
- No record of any prescription for the drugs being compared during the 12 months (+30 days) preceding the index date, i.e.,
  - For the primary comparison of initiation of empagliflozin versus DPP4i, patients will not have any prescription for empagliflozin/any SGLT2i or any DPP4i during the preceding 12 months (+30 days).
  - For the comparison of initiation of SGLT2i versus GLP1RA, patients will not have any prescription for any SGLT2i or any GLP1RA during the preceding 12 months (+30 days).

Patients will be excluded if they meet any of the following criteria:

- Aged <18 years on the first prescription date of the qualifying prescription,
- Pre-existing diagnosis of T1DM during the 12 months before the index date,
- Having a disqualifying diagnosis during the 12 months before the index date, defined as having at least one of the following: eGFR<30, dialysis, polycystic kidney disease or a kidney transplant,
- <12 months of available data before the index date, and/or no complete history of drug dispensations/other records of drug use during this period, defined as not having at least 1 ambulatory visit and at least 1 medication prescription during the preceding 12 months, and
- Missing or ambiguous data on serum creatinine in the 12 months prior to the index date or sex.

Patients will enter the study cohort on the date of their incident prescription for empagliflozin, SGLT2i, or comparator drug (baseline date) during 2015 – 2020. Baseline data will be determined from records at the baseline encounter, and from other health system encounters up to 12 months prior to baseline. Follow-up data (relevant medication prescriptions, measurements, and records for determining outcomes) will be collected until 31 December 2021 (study end date), but outcomes will be censored at 2 years after index date or end of data collection, if earlier.

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

**BI Study Number 1245-0228** 

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7.4.2 Preliminary patient counts

Preliminary estimates from 18 datamarts indicate a potential total sample size around 200,000 patients. The table below conveys estimated patient numbers obtained during the Study Specific Data Characterization (SSDC) and some of the following criteria will be modified for the final analytic query. Additionally, criteria 7 and alternative criteria 7 will be applied jointly as required exclusion criteria.

| Sequence | Inclusion/Exclusion Criteria | Estimated Sample<br>Size | % of Starting Cohort |
|---|---|---|---|
| 1 | Any record of prescription for empagliflozin, any SGLT2i, any DPP4 inhibitor, or any GLP1 use between 2014 and 2020 | 499671 | 100.0 |
| 2 | Adult >= 18 at date when criterion 1 is met | 499224 | 99.9 |
| 3 | Having a diagnosis of type 2 diabetes in 24 months before (including) the index date, based on ICD codes or other available data. | 337416 | 67.5 |
| 4 | Exclude pre-existing diagnosis of T1DM during the 12 months before the index date | 331350 | 66.3 |
| 5 | Exclude if record of any prescription for SGLT2i during the 12 months preceding the index date | 331096 | 66.3 |
| 6 | Exclude having one of the following during the 12 months before the index date: dialysis, polycystic kidney disease or a kidney transplant | 324970 | 65.0 |
| 7 | Exclude no record of ambulatory (AV) or telehealth (TH) visit during the 12 months before the index date | 261298 | 52.3 |
| 8 | Exclude missing serum creatinine in 24 months before the index date | 214810 | 43.0 |
| 9 | Exclude ambiguous or missing gender | 214806 | 43.0 |
| | Total patients identified above | 214806 | |
| Alternative Criteria | | | |
| 7 | Exclude no record of any prescription during the 12 months before the index date | 259772 | 52.0 |
| 8 | Exclude missing serum creatinine in 24 months before the index date | 211761 | 42.4 |

**Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

(NIS)

## BI Study Number 1245-0228

c39712001-02


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Sequence | Inclusion/Exclusion Criteria | Estimated Sample<br>Size | % of Starting Cohort |
|---|---|---|---|
| 9 | Exclude ambiguous or missing gender | 211758 | 42.4 |
| | Total patients identified above | 211758 | |

#### 7.5 **STUDY VISITS**

#### 7.5.1 Baseline period (lookback period)

Patients are required to have activity in their respective EHR at least 12 months prior to initiation of empagliflozin, SGLT2i or a comparator drug (index date). The look-back period is defined as 12 months prior to the index date and includes the index date. The look-back period was specified to confirm new medication use (i.e., having a first prescription for empagliflozin, any SGLT2i, DPP4i, or GLP1RA without use of these medications in the prior 12 months) and describe baseline parameters, such as prior medical history and medications. (See table 1 below for details related to timing of variable assessment).

Patients will enter the study cohort on the date of their incident prescription for empagliflozin, other SGLT2i, or comparator drug (baseline date) during 1 January 2015 – 31 December 2020. Baseline data will be determined from records at the baseline encounter, and from other health system encounters up to 12 months prior to baseline (see Table 1 for specific look back periods according to variable type).

Table 1 Variable types, assessment timeframes, and lookback periods

| Variable Type | 1 Year Prior to<br>Baseline | Baseline | +/- 3<br>months<br>from<br>baseline | +/- 30<br>days<br>from<br>baseline | Post baseline |
|---|---|---|---|---|---|
| Demographics | | X | | | |
| Medication<br>Prescriptions | X | X | | | X |
| Medical History | X | | | | |
| Labs | | | X | | X |
| Vitals | | | | X | |
| Hospitalization<br>Events | | | | | X |
| Death | | | | | X |


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8. VARIABLES

#### 8.1 EXPOSURES

Primary exposure:

- Main comparison:
  - Incident prescription order of empagliflozin without prior use of any SGLT2i or DPP4 inhibitors
  - Incident prescription order of any DPP4 inhibitor without prior use of any DPP4 inhibitor or any SGLT2i
- Secondary comparison:
  - Incident prescription order of any SGLT2i without prior use of SGLT2i or GLP1RA
  - Incident prescription order of any GLP1RA without prior use of any GLP1RA or SGLT2i

A modified As-Treated (AT) approach will be used for all analyses. Patients will be included in their incident prescription cohort with censoring occurring for the following reasons:

- Empagliflozin user has new prescription for a different SGLT2i during follow-up
- Empagliflozin [SGLT2i] user has new prescription for the comparator drug of interest during follow-up
- DPP4i or GLP1RA user has new prescription for any SGLT2i during follow-up
- No additional prescription for the incident drug has been written in the 1 year (+30 days) since the last observed prescription

This modified approach will be used due to inconsistencies across sites in completeness of the discontinuation dates in the prescription data and not having claims/fill data to supplement the written orders. We will assume a patient is on their initial prescription unless the criteria above have been met.

To better understand potential limitations of this modified AT approach, a feasibility assessment will be performed once the initial data queries are performed to quantify the availability of more detailed prescribing information (e.g., number of fills, number of pills, prescription end dates) across participating healthcare sites. If feasibility is determined by the investigative team, sensitivity analyses will be performed including sites with more complete prescribing information examining all primary and secondary outcomes (See Section 11.5).

The intention-to-treat (ITT) approach will be used as a sensitivity analysis for the primary and secondary comparisons of the primary outcome. In this ITT analysis, follow-up will not be censored when a patient switches to, or adds, treatment with a different agent, or does not receive a follow-up prescription for the incident drug.


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Primary subgroup of interest: diabetic kidney disease (DKD)

• DKD will be defined using diagnosis codes and laboratory values based on records at the index encounter and from other health system encounters up to 12 months prior to index prescription. Analyses will be performed overall and within subgroups of DKD (DKD and no DKD prior to or at baseline).

## 8.1.1 Study medications

For this study, eligible patients will be identified by the occurrence of a prescription for the following study medications of interest (index medications):

## Empagliflozin:

- Jardiance (empagliflozin)
- Synjardy (empagliflozin/metformin hydrochloride)

#### Other SGLT2i:

- Invokana (canagliflozin)
- Forxiga (dapagliflozin)
- Steglatro (ertugliflozin)

#### DPP4i:

- Januvia (sitagliptin)
- Galvus (vildagliptin)
- Onglyza (saxagliptin)
- Vipidia (alogliptin)
- Trajenta (linagliptin)
- Janumet (sitagliptin/metformin hydrochloride)
- Eucreas (vildagliptin/metformin hydrochloride)
- Kombiglyze (saxagliptin/metformin hydrochloride)
- Vipdomet (alogliptin/metformin hydrochloride)
- Jentadueto (linagliptin/metformin hydrochloride)

#### GLP1RA:

- Trulicity (dulaglutide)
- Tanzeum (albiglutide)
- Byetta (exenatide)
- Bydureon (exenatide once weekly)
- Victoza (liraglutide)

If additional SGLT2i, DPP4i or GLP1RA drugs are marketed in US during the study period, they will be added to the comparator group.

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

**BI Study Number 1245-0228** 

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Fixed-dose combinations of empagliflozin inhibitors with DPP-4 inhibitors, such as Glyxambi (empagliflozin/linagliptin), will not be included in either study cohort.

## 8.1.2 Operational definitions on how to identify each of the index medication cohorts

For index medication determination, we first select all patients with prescriptions for empagliflozin, any SGLT2i, any DPP4i, or any GLP1RA between 1 January 2015 and 31 December 2020. The first prescription for a participant during the study period will be identified as the index medication. The details for empagliflozin initiators are provided in **Figure 1** and all other drugs follow the same approach.



Figure 1 Consort diagram of study population, the application of inclusion and exclusion criteria, and the resulting study cohorts

#### 8.1.3 Definition of censored follow-up end

The primary analyses for the study will be conducted utilizing a modified "as-treated" approach.

Follow-up starts from the day after the index date until the first of the following qualifying events has been met:

• First occurrence of outcome of interest

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Death
- 2 years following the index prescription
- End of query specific study period (December 31, 2021)
- Empagliflozin user starts a DPP4i or other type of SGLT2i, or if a DPP4i user starts any SGLT2i
  - o SGLT2i user starts a GLP1RA, or a GLP1RA user starts any SGLT2i
- No observed prescriptions for the index drug within 1 year (+30 days) from the last observed prescription

If it is not a treatment line comparator, patients are allowed to add a non-incretin/non-SGLT2i hypoglycemic agent to their index therapy and can also switch to non-incretin/non-SGLT2i hypoglycemic agents.

**Intention-to-treat sensitivity analysis**: Follow-up will <u>not</u> be censored at the time of a drug switch or add-on or lack of follow-up prescription, i.e., the criterion of ending follow-up with the switch/add-on date will not be applied for this analysis.

**Discontinuation sensitivity analysis #1**: Follow-up will be censored similar to that of the modified AT approach with the final censoring criterion changed to:

• No observed prescriptions for the index drug within 6 months (+30 days) from the last observed prescription

**Discontinuation sensitivity analysis #2**: In sites where more complete prescribing data are available, follow-up will be censored similar to that of the modified AT approach with the final censoring criterion defined by drug exposure, which will be estimated as follows:

A supply, indicating the duration of exposure after a prescription, will be defined for each prescription based on the amount prescribed. Duration of exposure will be estimated based on a combination of prescribing variables potentially populated by sites in the Common Data Model (i.e. days supply, number of pills (quantity) ordered, dose frequency, and number of refills, start date, end date).

The duration of the supply in days (exposure period) will be derived as: duration = (days supply) \* (refills + 1). If number of refills is missing then we will assume no refills.

If days supply is missing then we will derive it as (end date - start date + 1) if these dates are available. If these dates are not available we will derive days supply as quantity / (number of doses per day), if these variables are available.

If a subsequent supply was prescribed before the previous supply has finished, the start of the subsequent supply will be shifted. For example, if a patient received the first supply for 60 days and a subsequent prescription record at day 50 for another 60 days, the duration of the two supplies combined is 50+10+60=120 days, after shifting the start of the second supply with 10 days for which the patient had supply in storage from the first supply. To avoid artificially long exposure periods, however, a subsequent supply can be shifted with a maximum of 14 days, which is considered a reasonable time for patients to receive a new

BI Study Number 1245-0228

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c39712001-02

prescription prior to the end of their current prescription. Further, a subsequent supply could not be shifted over the grace period (GP).

A GP for 100% of the duration of the most recent supply will be included in the exposure period to account for uncertainty related to actual drug use patterns. Overlapping supplies and GPs will be combined as exposure periods. The GP will be defined from the most recent prescription. In the above example on two overlapping supplies with 60 days, totaling in 120 days, the GP is 60 days (100% of the most recent supply), which implies the total exposure period in this example is 50+10+60+60=180 days.

The discontinuation will be defined as the date of ending the GP.

If there is a gap between subsequent prescriptions of more than the GP (e.g., start date of subsequent prescription is more than GP after the end date of the previous prescription), then the drug will be considered as discontinued GP days after the end of the first series of prescriptions.

A traditional 'as-treated'(AT) approach will be utilized in these sensitivity analyses. This means that the follow-up will be censored at discontinuation of continuous exposure, or switching to a comparator drug, and that the outcomes related to effectiveness, and safety, will be observed until the end of the first continuous exposure to a study drug or switching.

## 8.2 OUTCOMES

Study outcomes will be defined based on diagnoses, tests, and procedures recorded in the outpatient visits or hospitalizations (International Statistical Classification of Diseases and Related Health Problems, 9<sup>th</sup> and 10<sup>th</sup> Revision [ICD-9 and ICD-10], Logical Observation Identifiers Names and Codes [LOINC] and Current Procedural Terminology [CPT]) during follow-up. Note that, unless otherwise specified, for hospitalizations, all diagnoses, i.e., primary and secondary discharge diagnoses, will be considered. Absence of any record with a diagnosis code for a condition will be taken to mean absence of the condition. Only the first event during follow-up for each outcome will be considered.

All-cause death will be ascertained using Datavant software. See <u>Section 9</u> Data Sources below for more information.

The list of all codes to be used in each database is available in Annex 4.

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 8.2.1 Primary outcomes

Table 2 Primary outcomes and definitions

| Outcome | Definition |
|---|---|
| Composite outcome including 40% decline in eGFR from baseline using 2 follow-up eGFR measurements Incident end-stage kidney disease (ESKD) All-cause death | 40% decline in eGFR from baseline: at least 2 measurements during follow-up of at least a 40% decline relative to baseline with 2 follow-up measurements separated by ≥ 28 days ESKD definition: at least 1 kidney transplant or ESKD diagnosis/procedure¹ or at least 2 dialysis diagnoses/procedures¹ separated by ≥ 28 days or eGFR<15 on 2 measurements separated by ≥ 28 days |

## 8.2.2 Secondary outcomes

Table 3 Secondary outcomes and definitions

| Outcomes | Definition <sup>1</sup> |
|---|---|
| Secondary Renal Effectiveness Outcomes | |
| Secondary outcome 1: 40% decline in eGFR from baseline using 2 follow-up eGFR measurements | Same as that used for the primary composite outcome |
| Secondary outcome 2: Incident end-stage kidney disease (ESKD) | As for ESKD definition from primary composite outcome |
| Secondary outcome 3: Dialysis | Incident dialysis, given dialysis in the 12 months preceding index date is a disqualifying diagnosis/procedure |
| Secondary outcome 4: Kidney transplant | Any procedure* associated with healthcare encounters, including hospitalizations and specialist outpatient and primary care encounters |
| Secondary CV Effectiveness Outcomes | |
| Secondary outcome 5: Composite outcome including - Hospitalization for heart failure - All-cause death | Any diagnosis* of heart failure associated with hospital admission, including inpatient and ED to inpatient encounters. |
| 711 Gause death | From death records provided by sites, supplemented with linkage using Datavant Software. |
| Secondary outcome 6: Hospitalization for heart failure | Any diagnosis* associated with hospital admission, including inpatient and ED to inpatient encounters |
| Secondary outcome 7: All-cause death | From death records provided by sites, supplemented with linkage using Datavant Software. |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Outcomes | Definition <sup>1</sup> |
|---|---|
| Secondary outcome 8: Composite outcome including - MI** - Stroke** - All-cause death - Coronary revascularization procedure | For MI and stroke, any inpatient diagnosis** associated with healthcare encounters, including inpatient and ED to inpatient For all-cause death, as for secondary outcome 7 |
| Secondary outcome 9: Composite outcome including - MI** - Stroke** - All-cause death | For MI and stroke, any inpatient diagnosis** associated with healthcare encounters, including inpatient and ED to inpatient For all-cause death, as for secondary outcome 7 |
| Secondary safety outcomes | |
| Secondary outcome 10: Diabetic ketoacidosis | Any diagnosis* associated with healthcare encounters in the inpatient setting |
| Secondary outcome 11: Severe hypoglycemia | Any diagnosis* associated with healthcare encounters in the inpatient or ED setting |
| Secondary outcome 12: Urinary tract cancer | Two or more diagnoses* associated with healthcare encounters within 2 months |
| Secondary outcome 13: Severe Urinary Tract Infections | Any diagnosis¹ associated with healthcare encounters in the inpatient or ED setting for: • Pyelonephritis (ICD-10 codes in Annex Table 5 • -6) • Urosepsis. Combination of diagnosis code for UTI and a diagnosis code for sepsis within 1 week (ICD-10 codes for sepsis in Annex Table 5-6, ICD-10 codes for UTI in Annex Table 5-8). • In order to rule out nosocomial infection, at least one of the following criteria will have to be present within 7 days prior to the hospital admission: • Prescription for an antimicrobial agent • Outpatient visit with a recorded diagnosis code for UTI or pyelonephritis Outpatient visit with a recorded diagnosis code for UTI or pyelonephritis |
| Secondary outcome 14: Acute kidney injury that requires dialysis | Any diagnosis* associated with inpatient healthcare encounters for AKI plus at least one inpatient encounter indicating dialysis within 28 days of the AKI encounter Two or more dialysis encounters separated by 28 or |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

## BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Outcomes | Definition <sup>1</sup> |
|---|---|
| | more days will not be counted as an event. |
| Secondary outcome 15: Genital Mycotic Infection | Any diagnosis associated with healthcare encounters, including hospitalizations and outpatient encounters, or prescription for fluconazole |

<sup>\*</sup>Detailed variable definitions for the outcomes will be defined based on ICD diagnosis and procedure codes and CPT codes;

\*\*As heart failure, MI and stroke are defined from diagnosis without death data, the outcomes include both fatal and non-fatal events.



#### 8.3 COVARIATES

Listed below are the variables that will be used as a descriptive variable or covariate in the proposed analyses. The table below includes the list of variable names, the source of the variable within the PCORnet CDM and the variable definition.

| Variable Name | Source Table | Definition |
|---|---|---|
| Age | DEMOGRAPHIC | Calculated from DOB variable in DEMOGRAPHIC table. |
| Sex | DEMOGRAPHIC | SEX |
| Race/ethnicity | DEMOGRAPHIC | RACE<br>HISPANIC |
| Site<br>Region | HARVEST | DATAMARTID |
| Quarter and year of study entry | PRESCRIBING | |
| Blood pressure | VITAL | DIASTOLIC<br>SYSTOLIC |
| BMI<br>Obesity/overweight | VITAL | ORIGINAL_BMI<br>HEIGHT<br>WEIGHT |
| Smoking history | VITAL | SMOKING |
| Death | DEATH | DEATH_DATE |
| Ace/ARB use Beta blocker use Calcium-channel blocker use | PRESCRIBING | RXNORM_CUI |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Variable Name | Source Table | Definition |
|---|---|---|
| Thiazide diuretics | | |
| Loop diuretics | | |
| Other diuretics | | |
| Finerenone | | |
| sMRAs | | |
| Nitrates | | |
| Other Hypertension drugs | | |
| Digoxin use | | |
| Anti-arrhythmics | | |
| COPD or asthma medications | | |
| ARNi use | | |
| Statin use | | |
| Other lipid-lowering drugs | | |
| Antiplatelet agents | | |
| Oral anticoagulants | | |
| Heparin and other low-<br>molecular weight heparins | | |
| Nonsteroidal anti- | | |
| inflammatory drugs | | |
| Oral corticosteroids | | |
| Bisphosphonates | | |
| Opioids | | |
| Antidepressants | | |
| Antipsychotics | | |
| Anticonvulsants | | |
| Benzodiazepines | | |
| Other anxiolytics or hypnotics | | |
| Dementia medications | | |
| Antiparkinsonian medications | | |
| Metformin use | | |
| Sulfonylureas use | | |
| Insulin use | | |
| Glitazones | | |
| Number of anti-diabetic drugs | | |
| Monotherapy | | |
| Fluconazole | | |
| Charlson Comorbidity Index | DIAGNOSIS | DX |
| components | PROCEDURE | PX |
| Diabetic nephropathy | | |
| Diabetic retinopathy | | |
| Diabetes with other | | |
| ophthalmic conditions or | | |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Variable Name | Source Table | Definition |
|---|---|---|
| ophthalmic procedures | | |
| Diabetic neuropathy | | |
| Diabetes with peripheral | | |
| circulatory disorders | | |
| Diabetic Foot | | |
| Lower extremity amputation | | |
| Skin infections | | |
| Foot ulcer | | |
| Erectile dysfunction | | |
| Hypoglycemia (Any and severe) | | |
| Hyperglycemia | | |
| Disorders of fluid electrolyte and acid-base balance | | |
| Diabetic ketoacidosis | | |
| Volume depletion | | |
| Hyperosmolar hyperglycemic non-ketotic syndrome | | |
| Diabetes with unspecified complication | | |
| Alcohol abuse or dependence | | |
| Drug abuse or dependence | | |
| Ischemic heart disease | | |
| Acute myocardial infarction | | |
| Old myocardial infarction | | |
| Unstable angina | | |
| Stable angina | | |
| Other chronic ischemic heart disease | | |
| Coronary revascularization (PCI and CABG) | | |
| Ischemic or hemorrhagic stroke | | |
| Ischemic stroke | | |
| Transient ischemic attack | | |
| Hemorrhagic stroke and other cerebrovascular disease | | |
| Heart failure | | |
| Peripheral arterial disease | | |
| Lower extremity | | |
| revascularization | | |
| Atrial fibrillation | | |
| Other cardiac dysrhythmia | | |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Variable Name | Source Table | Definition |
|---|---|---|
| Other cardiovascular disease | | |
| Hypertension | | |
| Hyperlipidemia | | |
| Edema | | |
| Acute kidney injury | | |
| Dialysis | | |
| Hypertensive nephropathy | | |
| Kidney or bladder stones | | |
| Genital mycotic infection | | |
| Urinary tract infections (Any and Complicated) | | |
| Urinary tract cancer | | |
| COPD | | |
| Asthma | | |
| Pulmonary hypertension | | |
| Obstructive sleep apnea | | |
| Pneumonia | | |
| Liver disease | | |
| Osteoarthritis | | |
| Other arthritis, arthropathies and musculoskeletal pain | | |
| Dorsopathies | | |
| Fractures | | |
| Falls | | |
| Osteoporosis | | |
| Disorders of thyroid gland | | |
| Depression | | |
| Anxiety | | |
| Sleep disorders | | |
| Dementia | | |
| Delirium | | |
| Psychosis | | |
| Kidney transplant | | |
| End-stage kidney disease | | |
| Cancer | | |
| Coronary Artery Disease | | |


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

## **BI Study Number 1245-0228**

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Variable Name | Source Table | Definition |
|--------------------------|---------------|-----------------|
| Baseline DKD status/eGFR | LAB_RESULT_CM | LAB_LOINC |
| HbA1c | | RESULT_NUM |
| Creatinine | | RESULT_MODIFIER |
| BUN | | RESULT_UNIT |
| Total cholesterol | | |
| LDL | | |
| HDL | | |
| Triglycerides | | |

#### Model covariates:

- Any baseline variable that has an ASMD>0.10 after performing weighting that the clinical team evaluates as necessary.

The variables listed below will either be included in the propensity score (PS) modeling for patient weighting and/or presented in descriptive analyses for the baseline variables but will not be included in PS modeling (as indicated):

| Covariate | Keep in PS Model | Keep in baseline table,<br>not in PS model |
|---|---|---|
| Demographics | • | |
| Age | X | |
| Sex | X | |
| Race | X | |
| Site | X | |
| Region | | X |
| Calendar time (Quarter and year of cohort entry) | X | |
| Combined comorbidity score | X (Charleston<br>Comorbidity index) | |
| Diabetes-related complications | | |
| Diabetic nephropathy | X | |
| Diabetic retinopathy | X | |
| Diabetes with other ophthalmic conditions or ophthalmic procedures | X | |
| Diabetic neuropathy | X | |
| Diabetes with peripheral circulatory disorders | X | |
| Diabetic Foot | X | |
| Lower extremity amputation | X | |
| Skin infections | X | |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Covariate | Keep in PS Model | Keep in baseline table,<br>not in PS model |
|---|---|---|
| Foot ulcer | X | |
| Erectile dysfunction | | X |
| Hypoglycemia | X | |
| Hyperglycemia | X | |
| Disorders of fluid electrolyte and acid-base balance | X | |
| Diabetic ketoacidosis | X | |
| Hyperosmolar hyperglycemic non-ketotic syndrome | X | |
| Diabetes with unspecified complication | X | |
| Diabetes Complication Severity Index | | X |
| Features of diabetes medication initiation and baseling | ne diabetes therapy | |
| No. antidiabetic drugs at cohort entry | X | |
| Monotherapy | | X |
| Concomitant initiation or current use of metformin | X | |
| Concomitant initiation or current use of sulfonylureas | X | |
| Concomitant initiation or current use of insulin | X | |
| Concomitant initiation or current use of GLP-1 RAs | X | |
| Concomitant initiation or current use of glitazones | X | |
| Lifestyle factors and comorbidities | | • |
| BMI | X | |
| Obesity | | X |
| Overweight | | X |
| Smoking | X | |
| Alcohol abuse or dependence | X | |
| Drug abuse or dependence | X | |
| Ischemic heart disease | X | |
| Acute myocardial infarction | X | |
| Old myocardial infarction | X | |
| Unstable angina | X | |
| Stable angina | X | |
| Other chronic ischemic heart disease | X | |
| Previous coronary revascularization | X | |
| Ischemic or hemorrhagic stroke | | X |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Covariate | Keep in PS Model | Keep in baseline table,<br>not in PS model |
|---|---|---|
| Ischemic stroke | X | |
| Transient ischemic attack | X | |
| Hemorrhagic stroke and other cerebrovascular disease | X | |
| Heart failure | X | |
| Peripheral arterial disease | X | |
| Lower extremity revascularization | X | |
| Atrial fibrillation | X | |
| Other cardiac dysrhythmia | X | |
| Other cardiovascular disease | X | |
| Hypertension | X | |
| Blood pressure | X | |
| Hyperlipidemia | X | |
| Edema | | X |
| Non-diabetic renal dysfunction | | X |
| Acute kidney injury | X | |
| Chronic kidney disease | | X |
| Chronic kidney disease stage 1-2 | | X |
| Chronic kidney disease stage 3+ or dialysis | | X |
| Hypertensive nephropathy | X | |
| Miscellaneous renal insufficiency | | X |
| Kidney or bladder stones | | X |
| Urinary tract infections | X | |
| COPD | X | |
| Asthma | X | |
| Pulmonary hypertension | X | |
| Obstructive sleep apnea | X | |
| Pneumonia | X | |
| Liver disease | X | |
| Osteoarthritis | | X |
| Other arthritis, arthropathies and musculoskeletal pain | | X |
| Dorsopathies | | X |
| Fractures | X | |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Covariate | Keep in PS Model | Keep in baseline table, not in PS model |
|---|---|---|
| Falls | X | |
| Osteoporosis | X | |
| Disorders of thyroid gland | | X |
| Depression | | X |
| Anxiety | | X |
| Sleep disorders | | X |
| Dementia | | X |
| Delirium | | X |
| Psychosis | | X |
| Medications | | |
| Angiotensin converting enzyme inhibitors or<br>Angiotensin II receptor blockers | X | |
| Beta-blockers | X | |
| Calcium-channel blockers | X | |
| Thiazide diuretics | X | |
| Loop diuretics | X | |
| Other diuretics | X | |
| Finerenone | X | |
| sMRAs | X | |
| Nitrates | X | |
| Other hypertension drugs | X | |
| Digoxin | X | |
| Anti-arrhythmics | X | |
| COPD or asthma medications | | X |
| Statins | X | |
| Other lipid-lowering drugs | X | |
| Antiplatelet agents | X | |
| Oral anticoagulants | X | |
| Heparin and other low-molecular weight heparins | X | |
| Nonsteroidal anti-inflammatory drugs | | X |
| Oral corticosteroids | X | |
| Other immunosuppressives | X | |

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Covariate | Keep in PS Model | Keep in baseline table,<br>not in PS model |
|---|---|---|
| Bisphosphonates | X | |
| Opioids | X | |
| Antidepressants | | X |
| Antipsychotics | | X |
| Anticonvulsants | | X |
| Benzodiazepines | | X |
| Other anxiolytics or hypnotics | | X |
| Dementia medications | | X |
| Antiparkinsonian medications | | X |
| Measures of healthcare utilization (in prior yea | nr) | |
| Hospitalization within prior 30 days | X | |
| Hospitalization during prior 31-365 days | X | |
| No. hospitalizations | X | |
| No. hospital days | X | |
| No. emergency department visits | X | |
| No. office visits | X | |
| Electrocardiogram | | X |
| No. electrocardiograms | | X |
| No. distinct medication prescriptions | | X |
| No. HbA1c tests ordered | X | |
| No. glucose tests ordered | X | |
| No. microalbuminuria tests ordered | X | |
| No. creatinine tests ordered | X | |
| No. BUN tests ordered | X | |
| No. lipid tests | X | |
| Laboratory test results <sup>‡</sup> (results and ordered [y | //n]) | · |
| HbA1c (%) | X | |
| eGFR | X | |
| Creatinine (mg/dl) | | X |
| BUN (mg/dl) | X | |
| Total cholesterol (mg/dl) | X | |
| LDL level (mg/dl) | X | |


## Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Covariate | Keep in PS Model | Keep in baseline table,<br>not in PS model |
|---|---|---|
| HDL level (mg/dl) | X | |
| Triglyceride level (mg/dl) | X | |

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c39712001-02

## 9. DATA SOURCES

BI Study Number 1245-0228

This study will utilize high-quality renal function laboratory data available in medical electronic health records from approximately 20 health systems in the US that have mapped their data to the PCORnet CDM. Sites meeting PCORnet data curation quality checks will be eligible to participate in this study. Sites will be approached for participation in this study based on an initial feasibility assessment to determine the extent and completeness of key data elements (renal laboratory data, prescription data, relevant medical diagnoses, and data from both inpatient and outpatient encounters). Death data will be ascertained from site records and augmented with de-identified encrypted linkage to external sources, which includes reported deaths from the government and commercial obituaries using Datavant Software.


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10. DATA MANAGEMENT AND SOFTWARE/TOOLS

#### 10.1 SOFTWARE/TOOLS

SAS version 9.4 will be utilized for the analytic query to sites, data processing at statistical analysis. R version 4.0.2 or higher may be used for analysis.

#### 10.2 HANDLING OF MISSING VALUES

Missing data (e.g., for demographics, vital signs, lab measures) will be excluded from denominators in descriptive summaries. For propensity score models, extent of missing covariate data will be evaluated and appropriate measures for covariates such as sex, BMI, and lab results will be taken. For diagnoses, procedures and medications, absence of a relevant code during the specified time window will be interpreted as 'no evidence'. For these factors we hope to avoid possible misclassification through appropriate eligibility criteria (e.g., restricting to patients with evidence of interaction within the health system).

## 10.3 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS

Upon assessment of the data, outliers may be truncated to the 1<sup>st</sup> and 99<sup>th</sup> percentiles for modelling purposes only. Outliers will be included as is in descriptive summaries.

We do not expect extensive inconsistencies in the data. In the event that there are inconsistencies in lab values collected on the same day, we will use the average value for a given lab type across all values on that day.

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 11. DATA ANALYSIS

#### 11.1 PHASED APPROACH

A 2-part, phased approach will be utilized to complete the following analyses. The first phase of the analysis will include creating the demographics tables (unweighted and weighted) and CONNECT-S plots (overall and in the DKD and non-DKD subgroups), descriptive analyses of the prescribing data, and aggregated outcomes data. This will allow us to evaluate the degree of continued imbalance after weighting, consistency of prescribing data across treatment groups, and whether there is adequate power to assess outcomes under the current definitions.

The second phase of the analysis will be the completion of remaining analyses, given the first phase produces adequate results for continuing.

## 11.2 PROPENSITY SCORE MODELS AND OVERLAP WEIGHTING

For each two-arm comparison, propensity score models will be built using a logistic model with the covariates of interest and all subgroup by covariate pairwise interactions. The outcome of interest is treatment group, with empagliflozin [or any SGLT2i] as the treatment group of interest and DPP4i [or GLP1RA] as the reference treatment. LASSO will be used to select covariates and interactions to include. The variables/interactions that are remaining in the LASSO model are then refit to a standard logistic regression in order to estimate the final propensity score (PS) estimates and calculate the overlap weights. This approach is known as "post-LASSO" and is implemented because effects/probabilities from the LASSO model would be biased due to shrinkage of the coefficient estimates. Post-LASSO logistic modelling will be used to create propensity scores and calculate overlap weights within the DKD and no DKD groups separately.

For each patient, the overlap weight is the predicted propensity that the patient received the treatment opposite from what they were initiated on. Patients on the reference treatment are given a weight equal to PS, and for patients on the treatment of interest, the overlap weight is 1-PS. For example, for the comparison of empagliflozin versus DPP4i initiation, a patient who was initiated on empagliflozin will receive a weight equal to (1-PS), where PS is the estimated propensity score for empagliflozin initiation, and a patient who was initiated on DPP4i is weighted by PS. No trimming is required due to the PS weights being bounded between 0 and 1. Analysis of outcomes is then performed on the reweighted population (see Section 11.2 for a description of the PS weighting approach).

Absolute standardized mean differences between groups will be calculated to evaluate the success of the PS overlap weighting. Additionally, CONNECT-S plots will be created to visually depict the success of the overlap weighting.

BI Study Number 1245-0228

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c39712001-02

#### 11.3 DESCRIPTIVE ANALYSES

Baseline characteristics will be presented separately for each comparison cohort identified in sections above, resulting in one set of tables for each 2-arm comparison. Characteristics will include demographics, medical history, lab values, and concomitant medications. Continuous variables will be summarized as mean (standard deviation), median [5<sup>th</sup> percentile, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, and 95<sup>th</sup> percentile] and minimum, maximum. Categorical variables will be presented as frequencies (%), as will any continuous variable that is further categorized.

Characteristics will be presented in the unweighted cohorts. Additionally, characteristics will be stratified by DKD status and drug comparators. The degree of imbalance in variables between comparator arms will be quantified with absolute standardized mean differences.

Baseline characteristics will also be presented in the reweighted populations. Distributions of covariates in the DKD and no DKD groups and further within subgroups of interest will be assessed using standardized mean differences. Absolute standardized mean differences will be visually depicted using the CONNECT-S plot. Absolute standardized mean differences should be below or at 0.10 across covariates and subgroups. Any differences above 0.10 will be reviewed by the PIs and statistical team. If imbalances are determined to be clinically meaningful (e.g., based on overall prevalence and potential impact on outcomes) then these variables will be included as covariates in outcomes models.

Additionally, descriptive information on prescribing data for the index drug [class] will be presented, overall and by treatment group. The degree of missingness will be presented for every data field. The number of refills will be presented as a categorical variable, with categories of 0, 1, 2, 3, and 4+. Days supply will be summarized as a continuous variable, using mean (standard deviation), median [5<sup>th</sup> percentile, 25<sup>th</sup> percentile, 75<sup>th</sup> percentile, and 95<sup>th</sup> percentile] and minimum, maximum. The number of prescriptions for the index drug [class] per person during the follow-up period will be presented as a categorical variable. For patients with more than 1 prescription for the index drug during follow-up, the following will be described: average time (in days) between prescriptions and average time (in days) between index prescription and last prescription. For patients who switch drug during follow-up, the average time between index prescription and start of a new drug [class] will be summarized. Time to drug switching will be visualized using cumulative incidence functions, stratified by index drug [class].

## 11.4 COMPARATIVE EFFECTIVENESS ANALYSES

## 11.4.1 Empagliflozin vs. DPP4i

The effect of empagliflozin compared to DPP4i on outcomes will be assessed using Cox proportional hazards (PH) models in a 2-arm comparison. The analysis will include all patients with a valid overlap weight and will be performed for overall and within DKD

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

subgroups, using the reweighted population. The main analysis will assess outcomes while patients remain on initial treatment.

Follow-up will start the day after the index date (date of initiation of empagliflozin or DPP4i) and will continue until the first occurrence of the outcome of interest, or end of study date (date of death, date of study end, 2 years after index date). For the main "as treated" analysis (see **Section 8.1.** for more details), follow up will be censored early if an empagliflozin user starts a DPP4i or other type of SGLT2i, or if a DPP4i user starts any SGLT2i. If an empagliflozin or DPP4i user initiates a GLP1RA, this will be adjusted for in the model using a time-dependent indicator variable that takes the value of 1 when drug is initiated. Additionally, follow-up will be censored early if there is no indication of a new prescription in the 12 months (+30 days) following the last observed prescription.

Incidence rates will be computed as the number of first events per 1000 patient years of follow-up. Analyses of time to first event will be performed using Cox proportional hazards models. Outcomes where death is a competing risk will be analyzed using cause-specific proportional hazards models, achieved by censoring follow-up at the time of death. All analyses will be adjusted for covariates that continue to be unbalanced after reweighting, with any additional covariates that might be of medical interest identified by the clinicians. Hazard ratios comparing empagliflozin to DPP4i with 95% confidence intervals and the adjusted p-value for superiority will be presented for all outcomes.

The proportional hazards assumption will be checked for the treatment group variable using weighted Schoenfeld residuals (zph option in SAS). If the PH assumption is majorly violated, appropriate next steps will be taken. Options for next steps include adding an interaction with time, leaving the variable as is, or performing a stratified analysis. Plots will be visually checked to make the determination of a "major violation". Due to a potentially large sample size, significance testing could produce spurious significant results.

Kaplan-Meier curves will be created for each outcome in the overall and DKD subgroups using the reweighted population. Kaplan-Meier curves will also be generated to summarize the cumulative incidence of treatment switching by comparator arm.

Additionally, the total number of heart failure hospitalizations and the rate of heart failure hospitalization per 1000 patient years will be presented. The average number of HF hospitalizations per patient will be reported, in addition to the median (Q1, Q3) number of hospitalizations.

#### 11.4.2 SGLT2i vs. GLP1RA

We expect a sample size of  $\sim 3,000$  patients per group will provide adequate power to detect a HR of 0.75 with an incidence rate of 46 events per 1,000 patient years in the GLP1RA group.

Comparative effectiveness analyses described in **Section 11.4** will be repeated in a secondary comparison cohort of initiators of any SGLT2i or GLP1RA. In this analysis, follow up will
Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228 c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

also be censored if a SGLT2i user starts a GLP1RA, or if a GLP1RA user starts any SGLT2i. If a SGLT2i or GLP1RA user initiates a DPP4 inhibitor; this will be adjusted for in the model. Additionally, follow-up will be censored if there is no indication of a new prescription in the 12 months (+30 days) following the last observed prescription.



BI Study Number 1245-0228

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c39712001-02



#### 11.6 SAFETY ANALYSIS

Please see **Section 11** for analyses related to safety outcomes. The safety outcomes in this study are being evaluated similarly to all other outcomes of interest.

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS) BI Study Number 1245-0228 c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 12. QUALITY CONTROL

Validation or quality control (QC) refers to establishing by objective evidence that requirements of programming tasks have been implemented correctly and completely. To ensure these requirements are met, internal and beta testing is performed for every query according to applicable standard operating procedures (SOP). Data quality checks will include evaluating variable distributions to identify extreme outliers, which will be handled with input from the clinical PI. Key variables will be evaluated for unusual patterns of missingness or distributions over time and by site.

A Study Specific Data Characterization (SSDC) query will also be deployed to the selected sites to confirm data availability, completeness, conformance to the CDM specifications and study feasibility prior to the final production query. The SSDC will provide descriptive statistics of the data that will allow for an early evaluation of variable distributions. These results can often provide insights for local institutions to refine their data, and possibly refresh prior to the final query.

Additionally, as part of general QC standards, SAS log files will be saved after each production run and inspected for errors and warnings after each run by the program author. Log files will be free from ERROR messages, and any WARNINGS or problematic NOTEs, such as those concerning uninitialized variables or multi-record merging, etc., should be investigated and, if allowed to remain, should be reviewed with the lead statistician, with input from the statistical advisor if needed.

The statistical advisor will review new statistical results before they are released to the internal team, or in parallel (if timelines necessitate), and will review programming specifications and/or code as requested by the lead statistician, or as needed based on an assessment of risk. The clinical PI will review new statistical results before they are released to the sponsor.


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

- 1. Fleurence, R. L. et al. Launching PCORnet, a national patient-centered clinical research network. J Am Medical Informatics Assoc Jamia 21, 578–582 (2014).
- 2. Schernthaner G, et al. Evidence from routine clinical practice: EMPRISE provides a new perspective on CVOTs. Cardiovasc Diabetol. 2019 Aug 31;18(1):115. doi: 10.1186/s12933-019-0920-3.

#### 13.2 UNPUBLISHED REFERENCES

None.


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 14. ANNEXES

#### ANNEX 1. LIST OF STANDALONE DOCUMENTS

| Number | Document reference number | Description | Date | Title |
|---|---|---|---|---|
| 1 | c39368586-01 | Study Protocol (V 1.0) | 30 June<br>2022 | Comparative cardiovascular and renal effectiveness and safety of Empagliflozin and other SGLT2i in patients with type 2 diabetes (T2D) with and without baseline kidney disease in the United States |
| 2 | c39368586-02 | Study Protocol (V 2.0) | 26May2023 | Comparative cardiovascular and renal effectiveness and safety of Empagliflozin and other SGLT2i in patients with type 2 diabetes (T2D) with and without baseline kidney disease in the United States |
| 2 | c39712001-01 | Statistical and<br>Epidemiological Analysis<br>Plan (V 1.0) | 8 July 2022 | Statistical and Epidemiological Analysis Plan (SEAP) for Non- Interventional Study (NIS) to compare cardiovascular and renal effectiveness and safety of Empagliflozin and other SGLT2i in patients with type 2 diabetes (T2D) with and without baseline kidney disease in the United States – Version 1.0 |
| 4 | NA | Data Management and<br>Review Plan | 18 July<br>2022 | Comparative cardiovascular and renal effectiveness and safety of Empagliflozin and other SGLT2i in patients with type 2 diabetes (T2D) with and without baseline kidney disease in the United States: Data Management and Review Plan |
| 5 | TBD | Study codelist | 15June2023 | 1245.0228 Empa DKD<br>Codelist Master with<br>Sources 28Jul2023 |


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### **ANNEX 2. PROPOSED TABLES AND FIGURES**

Table 1a: Unweighted Baseline Characteristics of the Primary Comparison Cohort Population = Empagliflozin and DPP4i initiators

| Characteristic | Overall | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP41<br>Initiators | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| Demographics | | | | |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| Age (yrs) | | | | x.xx |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5th, 95th percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| Female sex | n (%) | n (%) | n (%) | x.xx |
| Race | | | | |
| Black | n (%) | n (%) | n (%) | x.xx |
| Other | n (%) | n (%) | n (%) | x.xx |
| White | n (%) | n (%) | n (%) | x.xx |
| Hispanic | n (%) | n (%) | n (%) | x.xx |
| Year of Index Prescription | | | | |
| 2015 | n (%) | n (%) | n (%) | x.xx |
| 2016 | n (%) | n (%) | n (%) | x.xx |
| 2017 | n (%) | n (%) | n (%) | x.xx |
| 2018 | n (%) | n (%) | n (%) | x.xx |
| 2019 | n (%) | n (%) | n (%) | x.xx |
| 2020 | n (%) | n (%) | n (%) | x.xx |
| Site Region | | | | |
| Northeast | n (%) | n (%) | n (%) | x.xx |
| North Central | n (%) | n (%) | n (%) | x.xx |
| South | n (%) | n (%) | n (%) | x.xx |
| West | n (%) | n (%) | n (%) | x.xx |
| Current smoker | n (%) | n (%) | n (%) | x.xx |
| Alcohol abuse/dependence | n (%) | n (%) | n (%) | x.xx |
| Drug abuse/dependence | n (%) | n (%) | n (%) | x.xx |
| Comorbidities | | | | |
| Charlson Comorbidity Index (Median [Q1, Q3]) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| Diabetes Complication Severity Index (Median, [Q1, Q3]) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| Ischemic heart disease | n (%) | n (%) | n (%) | x.xx |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| Hypertension | n (%) | n (%) | n (%) | x.xx |
| Hyperlipidemia | n (%) | n (%) | n (%) | x.xx |
| Heart Failure | n (%) | n (%) | n (%) | x.xx |
| MI | n (%) | 0 (0%) | n (%) | x.xx |
| Acute | n (%) | n (%) | n (%) | x.xx |
| History of | n (%) | n (%) | n (%) | x.xx |
| Unstable Angina | n (%) | n (%) | n (%) | x.xx |
| Stable Angina | n (%) | n (%) | n (%) | x.xx |
| Coronary Revascularization | n (%) | 0 (0%) | n (%) | x.xx |
| CAD | n (%) | n (%) | n (%) | x.xx |
| Ischemic Stroke | n (%) | 0 (0%) | n (%) | x.xx |
| Hemorrhagic Stroke | n (%) | n (%) | n (%) | x.xx |
| TIA | n (%) | n (%) | n (%) | x.xx |
| PAD | n (%) | n (%) | n (%) | x.xx |
| Atrial fibrillation | n (%) | n (%) | n (%) | x.xx |
| Other cardiac dysrhythmia | n (%) | n (%) | n (%) | x.xx |
| Edema | n (%) | n (%) | n (%) | x.xx |
| Cancer | n (%) | n (%) | n (%) | x.xx |
| Acute kidney injury | n (%) | n (%) | n (%) | x.xx |
| Chronic kidney disease | n (%) | n (%) | n (%) | x.xx |
| Stage 1-2 | n (%) | n (%) | n (%) | x.xx |
| Stage 3+ or dialysis | n (%) | n (%) | n (%) | x.xx |
| Hypertensive nephropathy | n (%) | n (%) | n (%) | x.xx |
| Kidney or bladder stones | n (%) | n (%) | n (%) | x.xx |
| Urinary tract infections | n (%) | n (%) | n (%) | x.xx |
| COPD | n (%) | n (%) | n (%) | x.xx |
| Asthma | n (%) | n (%) | n (%) | X.XX |
| Pulmonary hypertension | n (%) | n (%) | n (%) | X.XX |
| Obstructive sleep apnea | n (%) | n (%) | n (%) | X.XX |
| Pneumonia | n (%) | n (%) | n (%) | X.XX |
| Liver disease | n (%) | n (%) | n (%) | x.xx |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| Osteoarthritis | n (%) | n (%) | n (%) | x.xx |
| Dorsopathies | n (%) | n (%) | n (%) | x.xx |
| Fractures | n (%) | n (%) | n (%) | x.xx |
| Falls | n (%) | n (%) | n (%) | x.xx |
| Osteoporosis | n (%) | n (%) | n (%) | x.xx |
| Disorders of thyroid gland | n (%) | n (%) | n (%) | x.xx |
| Depression | n (%) | n (%) | n (%) | x.xx |
| Anxiety | n (%) | n (%) | n (%) | x.xx |
| Sleep disorders | n (%) | n (%) | n (%) | x.xx |
| Dementia | n (%) | n (%) | n (%) | x.xx |
| Delirium | n (%) | n (%) | n (%) | X.XX |
| Psychosis | n (%) | n (%) | n (%) | x.xx |
| <b>Diabetes Related Complications</b> | | | | |
| Diabetic nephropathy | n (%) | n (%) | n (%) | X.XX |
| Diabetic retinopathy | n (%) | n (%) | n (%) | X.XX |
| Diabetes with other ophthalmic conditions or ophthalmic procedures | n (%) | n (%) | n (%) | x.xx |
| Diabetic neuropathy | n (%) | n (%) | n (%) | X.XX |
| Diabetes with peripheral circulatory disorders | n (%) | n (%) | n (%) | x.xx |
| Diabetic Foot | n (%) | n (%) | n (%) | X.XX |
| Lower extremity amputation | n (%) | n (%) | n (%) | X.XX |
| Skin infections | n (%) | n (%) | n (%) | X.XX |
| Foot ulcer | n (%) | n (%) | n (%) | x.xx |
| Erectile dysfunction | n (%) | n (%) | n (%) | x.xx |
| Hypoglycemia | n (%) | n (%) | n (%) | x.xx |
| Hyperglycemia | n (%) | n (%) | n (%) | X.XX |
| Disorders of fluid electrolyte and acid-<br>base balance | n (%) | n (%) | n (%) | x.xx |
| Diabetic ketoacidosis | n (%) | n (%) | n (%) | x.xx |
| Hyperosmolar hyperglycemic non-<br>ketotic syndrome | n (%) | n (%) | n (%) | x.xx |
| Diabetes with unspecified complication | n (%) | n (%) | n (%) | x.xx |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| Labs and Vitals | | | | |
| SBP – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | x.xx |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| DBP – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | x.xx |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| BMI – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | x.xx |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| Overweight | n (%) | n (%) | n (%) | x.xx |
| Obesity | n (%) | n (%) | n (%) | x.xx |
| Serum creatinine – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | x.xx |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| eGFR – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | x.xx |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | XX, XX | xx, xx | |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| Albuminuria – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | X.XX |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| BUN – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | X.XX |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| HbA1c - N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | X.XX |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| $Total\ Cholesterol-N\ (\%)$ | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | X.XX |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| LDL – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | X.XX |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| HDL – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | x.xx |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| Triglycerides – N (%) | n (%) | n (%) | n (%) | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | X.XX |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | |
| Min, Max | xx, xx | xx, xx | xx, xx | |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | x.xx |
| <b>Medication History</b> | | | | |
| ACE inhibitors or ARBs | n (%) | n (%) | n (%) | X.XX |
| Beta blockers | n (%) | n (%) | n (%) | x.xx |
| Calcium-channel blockers | n (%) | n (%) | n (%) | x.xx |
| Thiazide diuretics | n (%) | n (%) | n (%) | x.xx |
| Loop diuretics | n (%) | n (%) | n (%) | x.xx |
| Other diuretics | n (%) | n (%) | n (%) | x.xx |
| Finerenone | n (%) | n (%) | n (%) | x.xx |
| sMRAs | n (%) | n (%) | n (%) | x.xx |
| Nitrates | n (%) | n (%) | n (%) | x.xx |
| Other hypertension drugs | n (%) | n (%) | n (%) | x.xx |
| Digoxin | n (%) | n (%) | n (%) | x.xx |
| Anti-arrhythmics | n (%) | n (%) | n (%) | x.xx |
| COPD or asthma medications | n (%) | n (%) | n (%) | X.XX |
| Other lipid-lowering drugs | n (%) | n (%) | n (%) | X.XX |
| Antiplatelet agents | n (%) | n (%) | n (%) | x.xx |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| Oral anticoagulants | n (%) | n (%) | n (%) | X.XX |
| Heparin and other low-molecular weight heparins | n (%) | n (%) | n (%) | x.xx |
| Nonsteroidal anti-inflammatory drugs | n (%) | n (%) | n (%) | X.XX |
| Oral corticosteroids | n (%) | n (%) | n (%) | x.xx |
| Other immunosuppressives | n (%) | n (%) | n (%) | x.xx |
| Bisphosphonates | n (%) | n (%) | n (%) | x.xx |
| Opioids | n (%) | n (%) | n (%) | x.xx |
| Antidepressants | n (%) | n (%) | n (%) | x.xx |
| Antipsychotics | n (%) | n (%) | n (%) | x.xx |
| Anticonvulsants | n (%) | n (%) | n (%) | x.xx |
| Benzodiazepines | n (%) | n (%) | n (%) | x.xx |
| Other anxiolytics or hypnotics | n (%) | n (%) | n (%) | x.xx |
| Dementia medications | n (%) | n (%) | n (%) | x.xx |
| Antiparkinsonian medications | n (%) | n (%) | n (%) | x.xx |
| ARNi | n (%) | n (%) | n (%) | x.xx |
| Statins | n (%) | n (%) | n (%) | x.xx |
| <b>Diabetes Medication History</b> | | | | |
| Monotherapy | n (%) | n (%) | n (%) | x.xx |
| Insulin | n (%) | n (%) | n (%) | x.xx |
| Metformin | n (%) | n (%) | n (%) | x.xx |
| Sulfonylureas | n (%) | n (%) | n (%) | x.xx |
| Glitazones | n (%) | n (%) | n (%) | x.xx |
| Empagliflozin | n (%) | n (%) | n (%) | x.xx |
| GLP1RA | n (%) | n (%) | n (%) | x.xx |
| DPP4 inhibitor | n (%) | n (%) | n (%) | X.XX |
| Other SGLT2i | n (%) | n (%) | n (%) | X.XX |
| Healthcare Utilization | | | | |
| Hospitalization within prior 30 days | n (%) | n (%) | n (%) | X.XX |
| Hospitalization during prior 31-365 days | n (%) | n (%) | n (%) | X.XX |
| No. hospitalizations | n (%) | n (%) | n (%) | X.XX |
| No. hospital days | n (%) | n (%) | n (%) | x.xx |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | Initiators | Absolute<br>Standardized<br>Mean<br>Difference |
|---|---|---|---|---|
| No. emergency department visits | n (%) | n (%) | n (%) | x.xx |
| No. office visits | n (%) | n (%) | n (%) | x.xx |
| Electrocardiogram | n (%) | n (%) | n (%) | x.xx |
| No. electrocardiograms | n (%) | n (%) | n (%) | x.xx |
| No. distinct medication prescriptions | n (%) | n (%) | n (%) | x.xx |

# Table 1b: Unweighted Baseline Characteristics of the Primary Comparison Cohort by DKD status Population = Empagliflozin and DPP4i initiators

| | Diabetic Kidney Disease | | No Diabetic Kidney Disease | | | |
|---|---|---|---|---|---|---|
| | Overall | Empagliflozir<br>Initiators | DPP4i<br>Initiators | Overall | Empagliflozir<br>Initiators | DPP4i<br>Initiators |
| Characteristic | (N=XXXX) | (N=XXXX) | (N=XXXX) | (N=XXXX) | (N=XXXX) | (N=XXXX) |
| Demographics | | | | | | |
| Age (yrs) | | | | | | |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Female sex | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Race | | | | | | |
| Black | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| White | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hispanic | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Year of Index Prescription | | | | | | |
| 2015 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| 2016 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| 2017 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| 2018 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| 2019 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| | Diabetic Kid | lney Disease | | No Diabetic Kidney Disease | | |
|---|---|---|---|---|---|---|
| Characteristic | Overall (N=XXXX) | Empagliflozir<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) |
| 2020 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Site Region | | | | | | |
| Northeast | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| North Central | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| South | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| West | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Current smoker | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Alcohol abuse/dependence | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Drug abuse/dependence | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Comorbidities | | | | | | |
| Charlson Comorbidity<br>Index (Median [Q1, Q3]) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Diabetes Complication<br>Severity Index (Median,<br>[Q1, Q3]) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Ischemic heart disease | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hypertension | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hyperlipidemia | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Heart Failure | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| MI | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Acute | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| History of | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Unstable Angina | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Stable Angina | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Coronary<br>Revascularization | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| CAD | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Ischemic Stroke | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hemorrhagic Stroke | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| TIA | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| PAD | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Atrial fibrillation | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| | Diabetic Kic | lney Disease | | No Diabetic | No Diabetic Kidney Disease | |
|---|---|---|---|---|---|---|
| Characteristic | Overall (N=XXXX) | Empagliflozir<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) |
| Other cardiac dysrhythmia | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Edema | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Cancer | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Acute kidney injury | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Chronic kidney disease | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Stage 1-2 | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Stage 3+ or dialysis | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hypertensive nephropathy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Kidney or bladder stones | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Urinary tract infections | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| COPD | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Asthma | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Pulmonary hypertension | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Obstructive sleep apnea | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Pneumonia | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Liver disease | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Osteoarthritis | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dorsopathies | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Fractures | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Falls | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Osteoporosis | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Disorders of thyroid gland | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Depression | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Anxiety | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Sleep disorders | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dementia | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Delirium | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Psychosis | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Diabetes Related<br>Complications | | | | | | |
| Diabetic nephropathy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| | Diabetic Kid | lney Disease | | No Diabetic | Kidney Diseas | e |
|---|---|---|---|---|---|---|
| Characteristic | Overall (N=XXXX) | Empagliflozir<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) |
| Diabetic retinopathy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Diabetes with other ophthalmic conditions or ophthalmic procedures | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Diabetic neuropathy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Diabetes with peripheral circulatory disorders | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Diabetic Foot | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Lower extremity amputation | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Skin infections | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Foot ulcer | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Erectile dysfunction | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hypoglycemia | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hyperglycemia | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Disorders of fluid electrolyte and acid-base balance | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Diabetic ketoacidosis | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hyperosmolar<br>hyperglycemic non-ketotic<br>syndrome | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Diabetes with unspecified complication | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Labs and Vitals | | | | | | |
| SBP – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| DBP – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| | Diabetic Kid | lney Disease | | No Diabetic | Kidney Diseas | e |
|---|---|---|---|---|---|---|
| Characteristic | Overall (N=XXXX) | Empagliflozir<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Overall (N=XXXX) | Empagliflozir<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| BMI – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Overweight | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Obesity | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Serum creatinine – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| N. Results in Prior Year<br>[Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| eGFR - N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| N. Results in Prior Year<br>[Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Albuminuria – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| N. Results in Prior Year<br>[Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| BUN – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| | Diabetic Kid | lney Disease | | No Diabetic | Kidney Diseas | e |
|---|---|---|---|---|---|---|
| Characteristic | Overall (N=XXXX) | Empagliflozir<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Overall (N=XXXX) | | DPP4i<br>Initiators<br>(N=XXXX) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| HbA1c – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| N. Results in Prior Year<br>[Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Total Cholesterol – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| N. Results in Prior Year<br>[Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| LDL - N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| N. Results in Prior Year<br>[Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| HDL – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| | Diabetic Kid | lney Disease | | No Diabetic Kidney Disease | | |
|---|---|---|---|---|---|---|
| Characteristic | Overall (N=XXXX) | Empagliflozir<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) |
| N. Results in Prior Year [Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| Triglycerides – N (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Mean (SD) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Median (Q1, Q3) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| Min, Max | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx | xx, xx |
| N. Results in Prior Year<br>[Median (Q1, Q3)] | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) | xx (xx, xx) |
| <b>Medication History</b> | | | | | | |
| ACE inhibitors or ARBs | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Beta blockers | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Calcium-channel blockers | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Thiazide diuretics | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Loop diuretics | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other diuretics | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Finerenone | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| sMRAs | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Nitrates | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other hypertension drugs | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Digoxin | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Anti-arrhythmics | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| COPD or asthma medications | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other lipid-lowering drugs | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Antiplatelet agents | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Oral anticoagulants | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Heparin and other low-<br>molecular weight heparins | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Nonsteroidal anti-<br>inflammatory drugs | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Oral corticosteroids | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| | Diabetic Kid | lney Disease | | No Diabetic | Kidney Diseas | se |
|---|---|---|---|---|---|---|
| Characteristic | Overall (N=XXXX) | Empagliflozir<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) | Overall (N=XXXX) | Empagliflozii<br>Initiators<br>(N=XXXX) | nDPP4i<br>Initiators<br>(N=XXXX) |
| Other immunosuppressives | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Bisphosphonates | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Opioids | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Antidepressants | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Antipsychotics | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Anticonvulsants | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Benzodiazepines | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other anxiolytics or hypnotics | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Dementia medications | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Antiparkinsonian medications | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| ARNi | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Statins | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Diabetes Medication<br>History | | | | | | |
| Monotherapy | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Insulin | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Metformin | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Sulfonylureas | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Glitazones | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Empagliflozin | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| GLP1RA | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| DPP4 inhibitor | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Other SGLT2i | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Healthcare Utilization | | | | | | |
| Hospitalization within prior 30 days | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Hospitalization during prior 31-365 days | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No. hospitalizations | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No. hospital days | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

Boehringer Ingelheim
Statistical and Enidemiological Analysis Plan (SEAP) for Nor


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | Diabetic Kid | ney Disease | | No Diabetic Kidney Disease | | |
|---|---|---|---|---|---|---|
| Characteristic | Overall (N=XXXX) | | Initiators | Overall | | DPP4i<br>Initiators<br>(N=XXXX) |
| No. emergency department visits | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No. office visits | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| Electrocardiogram | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No. electrocardiograms | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| No. distinct medication prescriptions | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |

Table 1c: Weighted Baseline Characteristics of the Primary Comparison Cohort Population = Empagliflozin and DPP4i initiators

Table 1d: Weighted Baseline Characteristics of the Primary Comparison Cohort by DKD status

**Population = Empagliflozin and DPP4i initiators** 

**Example Figure 1a: CONNECT-S Plot for the Primary Comparison Cohort, overall and by DKD status** 

**Population = Empagliflozin and DPP4i initiators** 



**BI Study Number 1245-0228** 

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# Table 1e: Prescribing Characteristics of the Primary Comparison Cohort Population = Empagliflozin and DPP4i initiators

| Characteristic | Overall (N=XXXX) | Empagliflozin<br>Initiators<br>(N=XXXX) | DPP4i<br>Initiators<br>(N=XXXX) |
|---|---|---|---|
| Missing Rx End Date (%) for Index Drug* | | | |
| Refills on Index Drug | | | |
| Missing | | | |
| 0 | | | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4+ | | | |
| Days Supply of Index Drug | | | |
| N Missing (%) | | | |
| Mean (SD) | | | |
| Median (Q1, Q3) | | | |
| 5 <sup>th</sup> , 95 <sup>th</sup> percentiles | | | |
| Min, Max | | | |
| Number of Index Drug Rx per patient | | | |
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4+ | | | |
| Time (days) between Rx for Index Drug [Mean (SD)] | 1 | | |
| Time (days) between first Rx and last Rx for Index Drug [Mean (SD)] | | | |
| Time (days) to switching [Mean (SD)] | | | |

empagliflozin group is supplied for empagliflozin prescriptions.

Figure 1b. Cumulative Incidence of Drug Switching During Follow-up, by Index Drug Population = Empagliflozin and DPP4i initiators

c39712001-02


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 2a: Unweighted Baseline Characteristics of the Secondary Comparison Cohort Population = SGLT2i and GLP1RA initiators

**Table 2b: Unweighted Baseline Characteristics of the Secondary Comparison Cohort by DKD status** 

**Population = SGLT2i and GLP1RA initiators** 

Table 2c: Weighted Baseline Characteristics of the Secondary Comparison Cohort Population = SGLT2i and GLP1RA initiators

**Table 2d: Weighted Baseline Characteristics of the Secondary Comparison Cohort by DKD status** 

**Population = SGLT2i and GLP1RA initiators** 

Figure 2a: CONNECT-S Plot for the Secondary Comparison Cohort, overall and by DKD status

**Population = SGLT2i and GLP1RA initiators** 

**Table 2e: Prescribing Characteristics of the Secondary Comparison Cohort Population = SGLT2i and GLP1RA initiators** 

Figure 2b. Cumulative Incidence of Drug Switching During Follow-up, by Index Drug Population = SGLT2i and GLP1RA initiators

c39712001-02


Table 3a: Effectiveness of Empagliflozin compared to DPP4i on Renal and CV Outcomes/ Population = Empagliflozin and DPP4i initiators

| | Empagliflozin | 1 | | DPP4i | | | | P-value |
|---|---|---|---|---|---|---|---|---|
| Outcome | Events<br>(PY1)<br>Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Events<br>(PY1)<br>Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Hazard<br>Ratio<br>(95% CI) | |
| Composite of 40% decline in eGFR, incident end-stage renal disease or all-cause death | | | | | | | | |
| Renal Effectiveness<br>Outcomes | | | | | | | | |
| 40% decline in eGFR | | | | | | | | |
| Incident end-stage renal disease | | | | | | | | |
| Dialysis | | | | | | | | |
| Kidney transplant | | | | | | | | |
| CV Effectiveness<br>Outcomes | | | | | | | | |
| Hospitalization for heart failure or all-cause death | | | | | | | | |
| Hospitalization for | | | | | | | | |


c39712001-02

| | Empagliflozin | | | DPP4i | | | | |
|---|---|---|---|---|---|---|---|---|
| Outcome | Events<br>(PY1)<br>Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Events<br>(PY1)<br>Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Hazard<br>Ratio<br>(95% CI) | P-value |
| heart failure | | | | | | | | |
| All-cause death | | | | | | | | |
| MI, stroke, all-cause<br>death, or coronary<br>revascularization | | | | | | | | |
| Safety Outcomes | | | | | | | | |
| Volume depletion | | | | | | | | |
| Diabetic ketoacidosis | | | | | | | | |
| Severe hypoglycemia | | | | | | | | |
| Urinary tract cancer | | | | | | | | |
| Complicated urinary tract infection | | | | | | | | |
| Acute kidney injury requiring dialysis | | | | | | | | |
| Genital mycotic infection | | | | | | | | |
| <b>Sensitivity Outcomes</b> | | | | | | | | |
| Composite of 40% decline in eGFR1, incident end-stage renal | | | | | | | | |

c39712001-02


| | Empagliflozin | | | DPP4i | | | | |
|---|---|---|---|---|---|---|---|---|
| Outcome | Events<br>(PY1)<br>Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Events<br>(PY1)<br>Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Hazard<br>Ratio<br>(95% CI) | P-value |
| disease or all-cause death | | | | | | | | |
| 40% decline in eGFR1 | | | | | | | | |
| Composite of 40% decline in eGFR, incident end-stage renal disease or all-cause death – ITT Approach | | | | | | | | |
| Composite of 40% decline in eGFR, incident end-stage renal disease or all-cause death – Discontinuation sensitivity analysis #1 | | | | | | | | |
| Composite of 40% decline in eGFR, incident end-stage renal disease or all-cause death – Traditional AT Approach (discontinuation sensitivity analysis #2) | | | | | | | | |
| Composite of 40% | | | | | | | | |

BI Study Number 1245-0228

Boehringer Ingelheim Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

c39712001-02


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| | Empagliflozin | | | DPP4i | | | | |
|---|---|---|---|---|---|---|---|---|
| | Events (PY1) | | | Events (PY1) | | | | |
| Outcome | Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Hazard<br>Ratio<br>(95% CI) | P-value |
| decline in eGFR, incident end-stage renal disease or all-cause death – eGFR excluded from PS models | | | | | | | | |

1For the primary outcome, eGFR decline is defined using 2 measurements. For the sensitivity outcome, only 1 measurement indicating decline will be required.

Table 3b: Effectiveness of Empagliflozin compared to DPP4i on Renal and CV Outcomes Population = Empagliflozin and DPP4i initiators with Diabetic Kidney Disease

Table 3c: Effectiveness of Empagliflozin compared to DPP4i on Renal and CV Outcomes Population = Empagliflozin and DPP4i initiators without Diabetic Kidney Disease

Figure 3x: Kaplan-Meier Event Curves Comparing Empagliflozin to DPP4i, overall and by DKD status Population = Empagliflozin and DPP4i initiatorsTable 4a: Effectiveness of SGLT2i compared to GLP1RA on Renal and CV Outcomes

**Population = SGLT2i and GLP1RA initiators** 

Table 4b: Effectiveness of SGLT2i compared to GLP1RA on Renal and CV Outcomes Population = SGLT2i and GLP1RA initiators with Diabetic Kidney Disease

Table 4c: Effectiveness of SGLT2i compared to GLP1RA on Renal and CV Outcomes Population = SGLT2i and GLP1RA initiators without Diabetic Kidney Disease

c39712001-02


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Figure 4x: Kaplan-Meier Event Curves Comparing SGLT2i to GLP1RA, overall and by DKD status Population = SGLT2i and GLPA1RA initiators

Table 5a: Baseline Characteristics of the Primary Comparison Cohort - Propensity Score Matching Population = Empagliflozin and DPP4i initiators

Table 5b: Baseline Characteristics of the Primary Comparison Cohort by DKD status – Propensity Score Matching Population = Empagliflozin and DPP4i initiators

Table 5c: Effectiveness of Empagliflozin compared to DPP4i on Renal and CV Outcomes - Propensity Score Matching Population = Empagliflozin and DPP4i initiators

Table 5d: Effectiveness of Empagliflozin compared to DPP4i on Renal and CV Outcomes - Propensity Score Matching Population = Empagliflozin and DPP4i initiators with Diabetic Kidney Disease

Table 5e: Effectiveness of Empagliflozin compared to DPP4i on Renal and CV Outcomes - Propensity Score Matching Population = Empagliflozin and DPP4i initiators without Diabetic Kidney Disease

Figure 5x: Kaplan-Meier Event Curves Comparing Empagliflozin to DPP4i, overall and by DKD status - Propensity Score Matching

**Population = Empagliflozin and DPP4i initiators** 


c39712001-02

c39712001-02


Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 7: Effectiveness of Empagliflozin compared to DPP4i on Renal and CV Outcomes in Subgroups - Population = Empagliflozin and DPP4i initiators

| | Empagliflozin | | | DPP4i | | | | |
|---|---|---|---|---|---|---|---|---|
| Outcome | Events (PY1) Median FU Time (Q1, Q3) | N at Risk | Incidence<br>Rate | Events (PY1)<br>Median FU<br>Time (Q1,<br>Q3) | N at Risk | Incidence<br>Rate | Hazard<br>Ratio<br>(95% CI) | Interaction<br>P-value |
| Sex | | | | | | | | |
| Male | | | | | | | | |
| Female | | | | | | | | |
| Age | | | | | | | | |
| <=65 | | | | | | | | |
| >65 | | | | | | | | |
| History of CV Events | | | | | | | | |
| Yes | | | | | | | | |
| No | | | | | | | | |
| History of HF Events | | | | | | | | |
| Yes | | | | | | | | |
| No | | | | | | | | |
| Concomitant metformin | | | | | | | | |
| Yes | | | | | | | | |
| No | | | | | | | | |


c39712001-02

| | Empagliflozin | | | DPP4i | | | | |
|---|---|---|---|---|---|---|---|---|
| Outcome | Events (PY1) Median FU Time (Q1, Q3) | N at Risk | Incidence<br>Rate | Events (PY1) Median FU Time (Q1, Q3) | N at Risk | Incidence<br>Rate | Hazard<br>Ratio<br>(95% CI) | Interaction P-value |
| eGFR (DKD Cohort only) | | | | | | | | |
| @30 | | | | | | | | |
| @40 | | | | | | | | |
| @50 | | | | | | | | |


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

**BI Study Number 1245-0228** 

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 3. REVIEWERS AND APPROVAL SIGNATURES

The NIS SEAP must be sent for review to the following individuals prior to approval.

| Reviewer | NIS involving BI product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi* | X | X | X |
| NIS Data Manager | X | X | X |
| TSTAT<br>(for NISnd only) | X | X | X |
| RWE CoE | X | X | |

<sup>\*</sup> When BI NIS lead is not TM Epi

**Study Title**: Comparative cardiovascular and renal effectiveness and safety of Empagliflozin and other SGLT2i in patients with type 2 diabetes (T2D) with and without baseline kidney disease in the United States

**Study Number: 1245.0228** 

**Protocol Version: 2.0** 

I herewith certify that I agree to the content of the study SEAP and to all documents

referenced in the study SEAP.





Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS) BI Study Number 1245-0228 c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

**ANNEX 4. CODELIST** 

BI Study Number 1245-0228

c39712001-02



BI Study Number 1245-0228

c39712001-02

DocuSign Envelope ID: 7BE3DD49-FB85-41C7-8861-1DAA3C5DD479

Boehringer Ingelheim
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

DX COVARIATE DX TIA TIA TA TO COVARIATE DX TIA TIA TIA TIA COVARIATE DX TIA TIA TIA COVARIATE DX TIA TIA TIA COVARIATE DX TIA TIA TIA COVARIATE DX TIA TIA TIA COVARIATE DX TIAS ANDINA UNITERALE ANDINA coverignment PROFESS

Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


DocuSign Envelope ID: 7BE3DD49-FB85-41C7-8861-1DAA3C5DD479

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


DocuSign Envelope ID: 7BE3DD49-FB85-41C7-8861-1DAA3C5DD479

### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


DocuSign Envelope ID: 7BE3DD49-FB85-41C7-8861-1DAA3C5DD479

## Boehringer Ingelheim Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


DocuSign Envelope ID: 7BE3DD49-FB85-41C7-8861-1DAA3C5DD479

## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


BI Study Number 1245-0228

Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

Proprietary confidential information © 2023 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


DocuSign Envelope ID: 7BE3DD49-FB85-41C7-8861-1DAA3C5DD479

#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  State of the state o

BI Study Number 1245-0228

c39712001-02


#### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


DocuSign Envelope ID: 7BE3DD49-FB85-41C7-8861-1DAA3C5DD479

### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

(NIS) Di Standar Nassach von 1245-0226

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


## Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the following of the followi

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


### Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


# Boehringer Ingelheim  State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


## **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| | CORONARY<br>REVASCULARIZATION, | | | | |
|---|---|---|---|---|---|
| PX_CABG | CABG (PX) | PXCH | 33510 | HEART ARTERY BYPASS, SINGLE | 33510 |
| PX_CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | 33511 | HEART ARTERY BYPASS , 2 GRAFTS | 33511 |
| PX CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | 33512 | HEART ARTERY BYPASS , 3 GRAFTS | 33512 |
| PX CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | 33513 | HEART ARTERY BYPASS , 4 GRAFTS | 33513 |
| | CORONARY REVASCULARIZATION, CABG (PX) | | | | |
| PX_CABG | CORONARY<br>REVASCULARIZATION, | PXCH | 33514 | HEART ARTERY BYPASS , 5 GRAFTS | 33514 |
| PX_CABG | CABG (PX) CORONARY REVASCULARIZATION, | PXCH | 33516 | HEART ARTERY BYPASS , 6 OR MORE GRAFTS COMBINED VEIN AND ARTERY HEART ARTERY | 33516 |
| PX_CABG | CABG (PX) | PXCH | 33517 | BYPASS | 33517 |
| PX_CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | 33518 | COMBINED VEIN AND ARTERY HEART ARTERY BYPASS, 2 GRAFTS | 33518 |
| PX CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | 33519 | COMBINED VEIN AND ARTERY HEART ARTERY BYPASS, 3 GRAFTS | 33519 |
| PX CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | 33521 | COMBINED VEIN AND ARTERY HEART ARTERY<br>BYPASS, 4 GRAFTS | 33521 |
| PX CABG | CORONARY REVASCULARIZATION, CABG (PX) | PXCH | 33522 | COMBINED VEIN AND ARTERY HEART ARTERY<br>BYPASS, 5 GRAFTS | 33522 |
| PX CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | 33523 | COMBINED VEIN AND ARTERY HEART ARTERY<br>BYPASS, 6 OR MORE GRAFTS | 33523 |
| PX CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | 33533 | HEART ARTERY BYPASS, SINGLE GRAFT | 33533 |
| _ | CORONARY<br>REVASCULARIZATION, | | | | |
| PX_CABG | CABG (PX) CORONARY REVASCULARIZATION, | PXCH | 33534 | HEART ARTERY BYPASS, 2 GRAFTS | 33534 |
| PX_CABG | CABG (PX) CORONARY | PXCH | 33535 | HEART ARTERY BYPASS, 3 GRAFTS | 33535 |
| PX_CABG | REVASCULARIZATION,<br>CABG (PX) | PXCH | 33536 | HEART ARTERY BYPASS, 4 OR MORE GRAFTS | 33536 |
| PX_CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | РХСН | S2205 | MINIMALLY INVASIVE DIRECT CORONARY ARTERY BYPASS SURGERY INVOLVING MINI-THORACOTOMY OR MINI-STERNOTOMY SURGERY, PERFORMED UNDER DIRECT VISION; USING ARTERIAL GRAFT(S), SINGLE CORONARY ARTERIAL GRAFT | S2205 |
| PX_CABG | CORONARY<br>REVASCULARIZATION,<br>CABG (PX) | PXCH | S2206 | MINIMALLY INVASIVE DIRECT CORONARY ARTERY BYPASS SURGERY INVOLVING MINI-THORACOTOMY OR MINI-STERNOTOMY SURGERY, PERFORMED UNDER DIRECT VISION; USING ARTERIAL GRAFT(S), TWO CORONARY ARTERIAL GRAFTS | S2206 |

Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| | | | | ELECTROCARDIOGRAM (ECG) 64 LEADS OR | |
|---|---|---|---|---|---|
| PX ECG | ELECTROCARDIOGRAM | PXCH | 0178T | GREATER WITH GRAPHIC PRESENTATION, ANALYSIS INTERPRETATION, AND REPORT | 0178T |
| PX_ECG | ELECTROCARDIOGRAM | PACH | 01781 | | 01781 |
| | | | | TRACING OF ELECTROCARDIOGRAM (ECG) 64 LEADS OR GREATER WITH GRAPHIC | |
| PX ECG | ELECTROCARDIOGRAM | PXCH | 0179T | PRESENTATION | 0179T |
| _ | | | | INTERPRETATION AND REPORT OF | |
| | | | | ELECTROCARDIOGRAM (ECG) 64 LEADS OR | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0180T | GREATER WITH GRAPHIC PRESENTATION | 0180T |
| | | | | REMOTE ANALYSIS OF ECG-DERIVED DATA WITH | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0206T | COMPUTER ASSESSMENT AND REPORT | 0206T |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0223T | ACOUSTIC ECG ANALYSIS | 0223T |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0224T | ACOUSTIC MULTIPLE INTERVAL ECG ANALYSIS | 0224T |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0225T | ACOUSTIC MULTIPLE INTERVAL ECG ANALYSIS | 0225T |
| | | | | EXTERNAL EKG RECORDING FOR MORE THAN 48 | |
| | | | | HOURS UP TO 21 DAYS WITH ANALYSIS, | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0295T | REPORT, REVIEW AND INTERPRETATION | 0295T |
| | | | | EXTERNAL EKG RECORDING FOR MORE THAN 48 | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0296T | HOURS UP TO 21 DAYS | 0296T |
| | | | | ANALYSIS AND REPORT OF EXTERNAL EKG | |
| | | | | RECORDING FOR MORE THAN 48 HOURS UP TO | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0297T | 21 DAYS | 0297T |
| | | | | REVIEW AND INTERPRETATION OF EXTERNAL | |
| | | | | EKG RECORDING FOR MORE THAN 48 HOURS UP | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 0298T | TO 21 DAYS | 0298T |
| | | | | ROUTINE EKG USING AT LEAST 12 LEADS | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93000 | INCLUDING INTERPRETATION AND REPORT | 93000 |
| | | | | ROUTINE ELECTROCARDIOGRAM (EKG) WITH | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93005 | TRACING USING AT LEAST 12 LEADS | 93005 |
| | | | | ROUTINE ELECTROCARDIOGRAM (EKG) USING | |
| | | | | AT LEAST 12 LEADS WITH INTERPRETATION AND | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93010 | REPORT | 93010 |
| | | | | TELEPHONIC TRANSMISSION OF | |
| | | | | POST-SYMPTOM ELECTROCARDIOGRAM | |
| | | | | RHYTHM STRIP(S), 24-HOUR ATTENDED | |
| 51/ 500 | | 51/01/ | | MONITORING, PER 30 DAY PERIOD OF TIME; | |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93012 | TRACING ONLY | 93012 |
| | | | | TELEPHONIC TRANSMISSION OF | |
| | | | | POST-SYMPTOM ELECTROCARDIOGRAM | |
| | | | | RHYTHM STRIP(S), 24-HOUR ATTENDED | |
| | | | | MONITORING, PER 30 DAY PERIOD OF TIME; | |
| DV FOC | EL ECTROCAPRIOCRAM | DVCII | 02044 | PHYSICIAN REVIEW WITH INTERPRETATION AND | 02044 |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93014 | REPORT ONLY | 93014 |
| DV ECC | EL ECTROCAPRIOCRAM | DVCH | 93025 | MEASUREMENT OF HEIGHT OF HEART BEATS ON EKG | 02025 |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93025 | | 93025 |
| | | | | TRACING OF ELECTRICAL ACTIVITY OF HEART | |
| PX ECG | ELECTROCARDIOGRAM | PXCH | 93040 | USING 1-3 LEADS WITH INTERPRETATION AND REPORT | 93040 |
| 1 X_LOO | LELOTROCARDIOGRAM | 1 XOII | 33040 | | 33040 |
| PX ECG | ELECTROCARDIOGRAM | PXCH | 93041 | TRACING OF ELECTRICAL ACTIVITY OF THE HEART USING 1-3 LEADS | 93041 |
| 17_200 | ELECTROCA (INDICOTO (IV) | 17,011 | 00041 | | 00041 |
| PX ECG | ELECTROCARDIOGRAM | PXCH | 93042 | INTERPRETATION AND REPORT OF ELECTRICAL ACTIVITY OF HEART USING 1-3 LEADS | 93042 |
| | LLCTITOOAIDIOOIVIII | 1 7.011 | 55042 | o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o o | 000-12 |
| | | | | HEART RHYTHM TRACING, ANALYSIS, AND | |
| | | | | INTERPRETATION OF 48-HOUR EKG, INCLUDES RECORDING, SCANNING ANALYSIS WITH | |
| PX ECG | ELECTROCARDIOGRAM | PXCH | 93224 | REPORT | 93224 |
| PX ECG | ELECTROCARDIOGRAM | PXCH | 93225 | HEART RHYTHM TRACING OF 48-HOUR EKG | 93225 |
| | | | | HEART RHYTHM ANALYSIS, INTERPRETATION | 1 |
| | | 1 | 1 | | |
| PX ECG | ELECTROCARDIOGRAM | PXCH | 93226 | AND REPORT OF 48-HOUR EKG | 93226 |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93226 | AND REPORT OF 48-HOUR EKG HEART RHYTHM TRACING, ANALYSIS, AND | 93226 |

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| PX ECG | ELECTROCARDIOGRAM | PXCH | 93228 | HEART RHYTHM TRACING, COMPUTER<br>ANALYSIS, AND INTERPRETATION OF<br>PATIENT-TRIGGERED EVENTS GREATER THAN<br>24-HOUR EKG UP TO 30 DAYS | 93228 |
|---|---|---|---|---|---|
| PX ECG | ELECTROCARDIOGRAM | PXCH | 93229 | HEART RHYTHM TRACING, COMPUTER ANALYSIS, PHYSICIAN PRESCRIBED TRANSMISSION OF PATIENT-TRIGGERED EVENTS GREATER THAN 24-HOUR EKG UP TO 30 DAYS | 93229 |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93230 | WEARABLE ELECTROCARDIOGRAPHIC RHYTHM DERIVED MONITORING FOR 24 HOURS BY CONTINUOUS ORIGINAL WAVEFORM RECORDING AND STORAGE WITHOUT SUPERIMPOSITION SCANNING UTILIZING A DEVICE CAPABLE OF PRODUCING A FULL MINIATURIZED PRINTOUT; INCLUDES RECORDING, MICROPROCESSOR-BASED ANALYSIS WITH REPORT, PHYSICIAN REVIEW AND INTERPRETATION | 93230 |
| PX_ECG | ELECTROCARDIOGRAM | РХСН | 93231 | WEARABLE ELECTROCARDIOGRAPHIC RHYTHM DERIVED MONITORING FOR 24 HOURS BY CONTINUOUS ORIGINAL WAVEFORM RECORDING AND STORAGE WITHOUT SUPERIMPOSITION SCANNING UTILIZING A DEVICE CAPABLE OF PRODUCING A FULL MINIATURIZED PRINTOUT; RECORDING (INCLUDES CONNECTION, RECORDING, AND DISCONNECTION) | 93231 |
| PX_ECG | ELECTROCARDIOGRAM | РХСН | 93232 | WEARABLE ELECTROCARDIOGRAPHIC RHYTHM DERIVED MONITORING FOR 24 HOURS BY CONTINUOUS ORIGINAL WAVEFORM RECORDING AND STORAGE WITHOUT SUPERIMPOSITION SCANNING UTILIZING A DEVICE CAPABLE OF PRODUCING A FULL MINIATURIZED PRINTOUT; MICROPROCESSOR-BASED ANALYSIS WITH REPORT | 93232 |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | 93233 | WEARABLE ELECTROCARDIOGRAPHIC RHYTHM DERIVED MONITORING FOR 24 HOURS BY CONTINUOUS ORIGINAL WAVEFORM RECORDING AND STORAGE WITHOUT SUPERIMPOSITION SCANNING UTILIZING A DEVICE CAPABLE OF PRODUCING A FULL MINIATURIZED PRINTOUT; PHYSICIAN REVIEW AND INTERPRETATION | 93233 |
| PX_ECG | ELECTROCARDIOGRAM | РХСН | 93235 | WEARABLE ELECTROCARDIOGRAPHIC RHYTHM DERIVED MONITORING FOR 24 HOURS BY CONTINUOUS COMPUTERIZED MONITORING AND NON-CONTINUOUS RECORDING, AND REAL-TIME DATA ANALYSIS UTILIZING A DEVICE CAPABLE OF PRODUCING INTERMITTENT FULL-SIZED WAVEFORM TRACINGS, POSSIBLY PATIENT ACTIVATED; INCLUDES MONITORING AND REAL-TIME DATA ANALYSIS WITH REPORT, PHYSICIAN REVIEW AND INTERPRETATION | 93235 |
| PX_ECG | ELECTROCARDIOGRAM | РХСН | 93236 | WEARABLE ELECTROCARDIOGRAPHIC RHYTHM DERIVED MONITORING FOR 24 HOURS BY CONTINUOUS COMPUTERIZED MONITORING AND NON-CONTINUOUS RECORDING, AND REAL-TIME DATA ANALYSIS UTILIZING A DEVICE CAPABLE OF PRODUCING INTERMITTENT FULL-SIZED WAVEFORM TRACINGS, POSSIBLY PATIENT ACTIVATED; MONITORING AND REAL-TIME DATA ANALYSIS WITH REPORT | 93236 |

Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| PX ECG | ELECTROCARDIOGRAM | РХСН | S0346 | ELECTROCARDIOGRAPHIC MONITORING UTILIZING A HOME COMPUTERIZED TELEMETRY STATION WITH AUTOMATIC ACTIVATION AND REAL-TIME NOTIFICATION OF MONITORING STATION, 24-HOUR ATTENDED MONITORING, INCLUDING RECORDING, MONITORING, RECEIPT OF TRANSMISSIONS, AND ANALYSIS; PER 24-HOUR PERIOD | S0346 |
|---|---|---|---|---|---|
| PX_ECG | ELECTROCARDIOGRAM | РХСН | S0347 | ELECTROCARDIOGRAPHIC MONITORING UTILIZING A HOME COMPUTERIZED TELEMETRY STATION WITH AUTOMATIC ACTIVATION AND REAL-TIME NOTIFICATION OF MONITORING STATION, 24-HOUR ATTENDED MONITORING, INCLUDING PHYSICIAN REVIEW AND INTERPRETATION; 24-HOUR PERIOD | S0347 |
| PX_ECG | ELECTROCARDIOGRAM | PXCH | S9025 | OMNICARDIOGRAM/CARDIOINTEGRAM | S9025 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 78.52 | INTERNAL FIXATION OF BONE WITHOUT FRACTURE REDUCTION, HUMERUS | 7852 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 78.53 | INTERNAL FIXATION OF BONE WITHOUT FRACTURE REDUCTION, RADIUS AND ULNA | 7853 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 78.55 | INTERNAL FIXATION OF BONE WITHOUT FRACTURE REDUCTION, FEMUR | 7855 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 79.01 | CLOSED REDUCTION OF FRACTURE WITHOUT INTERNAL FIXATION, HUMERUS | 7901 |
| PX FRACTURE | FRACTURES (PX) | PX09 | 79.02 | CLOSED REDUCTION OF FRACTURE WITHOUT INTERNAL FIXATION, RADIUS AND ULNA | 7902 |
| PX FRACTURE | FRACTURES (PX) | PX09 | 79.05 | CLOSED REDUCTION OF FRACTURE WITHOUT INTERNAL FIXATION, FEMUR | 7905 |
| PX FRACTURE | FRACTURES (PX) | PX09 | 79.11 | CLOSED REDUCTION OF FRACTURE WITH INTERNAL FIXATION, HUMERUS | 7911 |
| PX FRACTURE | FRACTURES (PX) | PX09 | 79.12 | CLOSED REDUCTION OF FRACTURE WITH INTERNAL FIXATION, RADIUS AND ULNA | 7912 |
| PX FRACTURE | FRACTURES (PX) | PX09 | 79.15 | CLOSED REDUCTION OF FRACTURE WITH INTERNAL FIXATION, FEMUR | 7915 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 79.21 | OPEN REDUCTION OF FRACTURE WITHOUT INTERNAL FIXATION, HUMERUS | 7921 |
| PX FRACTURE | FRACTURES (PX) | PX09 | 79.22 | OPEN REDUCTION OF FRACTURE WITHOUT INTERNAL FIXATION, RADIUS AND ULNA | 7922 |
| _ | | PX09 | 79.25 | OPEN REDUCTION OF FRACTURE WITHOUT INTERNAL FIXATION, FEMUR | 7925 |
| PX_FRACTURE | FRACTURES (PX) | | | OPEN REDUCTION OF FRACTURE WITH<br>INTERNAL FIXATION, HUMERUS | |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 79.31 | OPEN REDUCTION OF FRACTURE WITH | 7931 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 79.32 | INTERNAL FIXATION, RADIUS AND ULNA OPEN REDUCTION OF FRACTURE WITH INTERNAL FIXATION. FEMUR | 7932 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 79.35 | DEBRIDEMENT OF OPEN FRACTURE SITE, | 7935 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 79.61 | DEBRIDEMENT OF OPEN FRACTURE SITE, | 7961 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 79.62 | RADIUS AND ULNA DEBRIDEMENT OF OPEN FRACTURE SITE, | 7962 |
| PX_FRACTURE | FRACTURES (PX) | PX09 | 79.65 | FEMUR INSERTION OF INTERNAL FIXATION DEVICE INTO | 7965 |
| PX_FRACTURE | FRACTURES (PX) | PX10 | 0PHC04Z | RIGHT HUMERAL HEAD, OPEN APPROACH INSERTION OF EXTERNAL FIXATION DEVICE INTO | 0PHC04Z |
| PX_FRACTURE | FRACTURES (PX) | PX10 | 0PHC05Z | RIGHT HUMERAL HEAD, OPEN APPROACH | 0PHC05Z |
| PX_FRACTURE | FRACTURES (PX) | PX10 | 0PHC06Z | INSERTION OF INTRAMEDULLARY INTERNAL<br>FIXATION DEVICE INTO RIGHT HUMERAL HEAD,<br>OPEN APPROACH | 0PHC06Z |
| PX_FRACTURE | FRACTURES (PX) | PX10 | 0PHC08Z | INSERTION OF LIMB LENGTHENING EXTERNAL FIXATION DEVICE INTO RIGHT HUMERAL HEAD, OPEN APPROACH | 0PHC08Z |

Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

States and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the Additional Study

State of the Additional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| | | Byou | | CLOSED TREATMENT OF GROWTH PLATE OR<br>BROKEN UPPER ARM BONE AT ELBOW WITH | |
|---|---|---|---|---|---|
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24535 | MANIPULATION | 24535 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24538 | INSERTION OF HARDWARE TO GROWTH PLATE OR BROKEN UPPER ARM BONE AT ELBOW, ACCESSED THROUGH THE SKIN | 24538 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24545 | OPEN TREATMENT OF GROWTH PLATE OR<br>BROKEN UPPER ARM BONE AT ELBOW | 24545 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24560 | CLOSED TREATMENT OF BROKEN UPPER ARM BONE AT SHOULDER | 24560 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24565 | CLOSED TREATMENT OF BROKEN UPPER ARM BONE AT SHOULDER WITH MANIPULATION | 24565 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24575 | OPEN TREATMENT OF BROKEN UPPER ARM BONE AT ELBOW | 24575 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24586 | OPEN TREATMENT OF BROKEN AND/OR DISLOCATED UPPER OR LOWER ARM BONES AT ELBOW | 24586 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 24587 | OPEN TREATMENT OF BROKEN AND/OR DISLOCATED UPPER OR LOWER ARM BONES AT ELBOW WITH IMPLANT | 24587 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 24620 | CLOSED TREATMENT OF BROKEN AND DISLOCATED FOREARM BONES AT ELBOW WITH MANIPULATION | 24620 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 24635 | OPEN TREATMENT OF BROKEN AND DISLOCATED FOREARM BONES AT ELBOW | 24635 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24650 | CLOSED TREATMENT OF BROKEN FOREARM<br>BONE AT ELBOW | 24650 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24655 | CLOSED TREATMENT OF BROKEN FOREARM (RADIUS) BONE AT THE ELBOW AREA ON THE OUTSIDE PART OF THE ARM WITH MANIPULATION | 24655 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24665 | OPEN TREATMENT OF THE FOREARM BONE ON THE THUMB SIDE OF THE FOREARM (RADIUS BONE) IN THE ELBOW REGION | 24665 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24666 | OPEN TREATMENT OF BROKEN FOREARM BONE AT ELBOW WITH PROSTHETIC REPLACEMENT | 24666 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24670 | CLOSED TREATMENT OF BROKE FOREARM BONE AT ELBOW | 24670 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 24685 | OPEN TREATMENT OF THE FOREARM BONE ON<br>THE SMALL FINGER SIDE OF THE FOREARM<br>(ULNA BONE) IN THE ELBOW REGION | 24685 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 25500 | CLOSED TREATMENT OF BROKEN FOREARM<br>BONE (RADIUS) AT THE MID PORTION ON THE<br>THUMB SIDE OF THE ARM WITHOUT<br>MANIPULATION | 25500 |
| | | | | CLOSED TREATMENT OF BROKEN FOREARM<br>BONE (RADIUS) AT THE MID PORTION ON THE | |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25505 | THUMB SIDE OF THE ARM WITH MANIPULATION OPEN TREATMENT OF THE SHAFT OF THE | 25505 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25515 | FOREARM BONE ON THE THUMB SIDE OF THE FOREARM (RADIUS BONE) | 25515 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25530 | CLOSED TREATMENT OF BROKEN FOREARM<br>BONE (ULNA) AT THE MID PORTION ON THE<br>SMALL FINGER SIDE OF THE ARM WITHOUT<br>MANIPULATION | 25530 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25535 | CLOSED TREATMENT OF BROKEN FOREARM<br>BONE (ULNA) AT THE MID PORTION ON THE<br>SMALL FINGER SIDE OF THE ARM WITH<br>MANIPULATION | 25535 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25545 | OPEN TREATMENT OF THE SHAFT OF THE FOREARM BONE ON THE SMALL FINGER SIDE OF THE FOREARM, ULNA BONE | 25545 |

Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| | | | | OLOGED TREATMENT OF BOTH FOREADM | |
|---|---|---|---|---|---|
| PX FRACTURE | FRACTURES (PX) | PXCH | 25560 | CLOSED TREATMENT OF BOTH FOREARM BONES (ULNA AND ULNA) AT THE MID PORTION WITHOUT MANIPULATION | 25560 |
| | | | | CLOSED TREATMENT OF BROKEN FOREARM | |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25565 | BONES WITH MANIPULATION | 25565 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25575 | OPEN TREATMENT OF BROKEN BOTH FOREARM BONES | 25575 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 25600 | CLOSED TREATMENT OF BROKEN FOREARM<br>(RADIUS) BONE AT THE WRIST AREA ON THE<br>THUMB SIDE OF THE WRIST WITHOUT<br>MANIPULATION | 25600 |
| TX_TTACTORE | TIVACTOREO (FX) | 1 XOII | 23000 | CLOSED TREATMENT OF BROKEN OR GROWTH | 25000 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25605 | PLATE SEPARATE OF FOREARM BONE AT WRIST<br>WITH MANIPULATION | 25605 |
| PX_FRACTURE | FRACTURES (PX) | РХСН | 25611 | PERCUTANEOUS SKELETAL FIXATION OF DISTAL RADIAL FRACTURE (EG, COLLES OR SMITH TYPE) OR EPIPHYSEAL SEPARATION, WITH OR WITHOUT FRACTURE OF ULNAR STYLOID, REQUIRING MANIPULATION, WITH OR WITHOUT EXTERNAL FIXATION | 25611 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 25620 | OPEN TREATMENT OF DISTAL RADIAL FRACTURE (EG, COLLES OR SMITH TYPE) OR EPIPHYSEAL SEPARATION, WITH OR WITHOUT FRACTURE OF ULNAR STYLOID, WITH OR WITHOUT INTERNAL OR EXTERNAL FIXATION | 25620 |
| | | | | CLOSED TREATMENT OF BROKEN FOREARM AT | |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 25650 | WRIST BONE | 25650 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27125 | PARTIAL REPLACEMENT OF THIGH BONE AT HIP JOINT WITH PROSTHESIS | 27125 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27130 | REPLACEMENT OF THIGH BONE AND HIP JOINT PROSTHESIS | 27130 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 27193 | CLOSED TREATMENT OF PELVIC RING FRACTURE OR DISLOCATION | 27193 |
| | | | | CLOSED TREATMENT OF PELVIC RING FRACTURE OR DISLOCATION WITH | |
| PX_FRACTURE<br>PX_FRACTURE | FRACTURES (PX) FRACTURES (PX) | PXCH | 27194<br>27200 | MANIPULATION UNDER ANESTHESIA CLOSED TREATMENT OF BROKEN TAILBONE | 27194<br>27200 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27200 | OPEN TREATMENT OF BROKEN TAILBONE | 27202 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 27215 | OPEN TREATMENT OF BROKEN BONES ON ONE SIDE OF PELVIS | 27215 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27216 | INSERTION OF HARDWARE TO BROKEN AND/OR DISLOCATED BONE ON ONE SIDE OF PELVIS, ACCESSED THROUGH THE SKIN | 27216 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27217 | OPEN TREATMENT OF FRACTURE AND/OR DISLOCATION OF PELVIS, ANTERIOR | 27217 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27218 | OPEN TREATMENT OF FRACTURE AND/OR DISLOCATION OF PELVIS, POSTERIOR | 27218 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27220 | CLOSED TREATMENT OF HIP SOCKET FRACTURES | 27220 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27222 | CLOSED TREATMENT OF HIP SOCKET FRACTURES WITH MANIPULATION | 27222 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27226 | OPEN TREATMENT OF HIP SOCKET FRACTURE WITH INSERTION OF HARDWARE | 27226 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27227 | OPEN TREATMENT OF FRACTURE OF FRONT OR BACK COLUMN OF HIP SOCKET OR ACROSS HIP SOCKET WITH INSERTION OF FIXATION HARDWARE | 27227 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 27228 | OPEN TREATMENT OF FRACTURE OF FRONT<br>AND BACK COLUMN OR WALL OF HIP SOCKET<br>WITH INSERTION OF FIXATION HARDWARE | 27228 |
| | , , | | | CLOSED TREATMENT OF UPPER THIGH BONE FRACTURE | 27230 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 27230 | | |

Boehringer Ingelheim

State and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| PX_FRACTURE | FRACTURES (PX) | PXCH | 27235 | INSERTION OF HARDWARE TO BROKEN THIGH<br>BONE, ACCESSED THROUGH THE SKIN | 27235 |
|---|---|---|---|---|---|
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27236 | OPEN TREATMENT OF BROKEN THIGH BONE<br>WITH INSERTION OF HARDWARE OR<br>PROSTHETIC REPLACEMENT | 27236 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27238 | CLOSED TREATMENT OF FRACTURE BELOW NECK OF UPPER THIGH BONE | 27238 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27240 | CLOSED TREATMENT OF FRACTURE BELOW NECK OF THIGH BONE (INTERTROCHANTERIC OR SUBTROCHANTERIC) WITH MANIPULATION | 27240 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27244 | SURGICAL TREATMENT OF BROKEN THIGH BONE WITH PLACE/SCREW IMPLANT | 27244 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27245 | SURGICAL TREATMENT OF BROKEN THIGH BONE WITH IMPLANT | 27245 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27246 | CLOSED TREATMENT OF BROKEN HIP,<br>TROCHANTER | 27246 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27248 | OPEN TREATMENT OF BROKEN THIGH BONE USING INTERNAL FIXATION | 27248 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27254 | OPEN TREATMENT OF FRACTURE AND TRAUMATIC DISLOCATION OF HIP SOCKET AND THIGH BONE | 27254 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27267 | CLOSED TREATMENT OF BROKEN HIP, AT THE JOINT | 27267 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 27268 | CLOSED TREATMENT OF FRACTURE OF UPPER PORTION AND HEAD OF THIGH BONE WITH MANIPULATION | 27268 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27269 | OPEN TREATMENT OF FRACTURE OF THIGH<br>BONE | 27269 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27500 | CLOSED TREATMENT OF THIGH BONE FRACTURE | 27500 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27501 | CLOSED TREATMENT OF BROKEN THIGH BONE, KNEE AREA, WITHOUT MANIPULATION | 27501 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27502 | CLOSED TREATMENT OF BROKEN THIGH BONE, MID-PORTION WITH MANIPULATION | 27502 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27503 | CLOSED TREATMENT OF BROKEN THIGH BONE, KNEE AREA, MANIPULATION | 27503 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27506 | OPEN TREATMENT OF BROKEN THIGH BONE, WITH IMPLANT | 27506 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27507 | OPEN TREATMENT WITH PLATE/SCREWS OF BROKEN THIGH BONE | 27507 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27508 | CLOSED TREATMENT OF BROKEN THIGH BONE,<br>LOWER END, WITHOUT MANIPULATION, INSIDE<br>OR OUTSIDE PORTION | 27508 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27509 | INSERTION OF HARDWARE TO STABILIZE<br>BROKEN THIGH BONE OR SEPARATED GROWTH<br>PLATE, ACCESSED THROUGH THE SKIN | 27509 |
| OV EDAOTUBE | | DVOL | 07540 | OPEN TREATMENT OF FRACTURE OF LOWER END OF THIGH BONE JUST ABOVE KNEE JOINT (SUPRACONDYLAR OR TRANSCONDYLAR | 07540 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | 27513 | FRACTURE OF FEMUR) OPEN TREATMENT OF FRACTURE OF ONE SIDE | 27513 |
| PX FRACTURE | FRACTURES (PX) | PXCH | 27514 | OF LOWER END OF THIGH BONE JUST ABOVE<br>KNEE JOINT (MEDIAL OR LATERAL CONDYLE<br>FRACTURE OF FEMUR) | 27514 |
| PX_FRACTURE | FRACTURES (PX) | PXCH | G0412 | OPEN TREATMENT OF ILIAC SPINE(S), TUBEROSITY AVULSION, OR ILIAC WING FRACTURE(S), UNILATERAL OR BILATERAL FOR PELVIC BONE FRACTURE PATTERNS WHICH DO NOT DISRUPT THE PELVIC RING INCLUDES INTERNAL FIXATION, WHEN PERFORMED | G0412 |
Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the following of the followi

BI Study Number 1245-0228

c39712001-02


### **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


### **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


#### **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


# **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| DV LOWED AND | LOWER EXTREMITY (LIMB) AMPUTATION | DVCII | 27504 | AMPUTATION OF THIGH THROUGH THIGH BONE WITH IMMEDIATE FITTING | 27504 |
|---|---|---|---|---|---|
| PX_LOWER_AMP | (PX) | PXCH | 27591 | WITH IMMEDIATE FITTING | 27591 |
| PX LOWER AMP | LOWER EXTREMITY<br>(LIMB) AMPUTATION<br>(PX) | PXCH | 27592 | AMPUTATION OF THIGH THROUGH THIGH BONE,<br>OPEN PROCEDURE | 27592 |
| | LOWER EXTREMITY<br>(LIMB) AMPUTATION | | | AMPUTATION OF THIGH THROUGH THIGH BONE, | |
| PX_LOWER_AMP | (PX) LOWER EXTREMITY | PXCH | 27594 | SECONDARY CLOSURE | 27594 |
| PX_LOWER_AMP | (LIMB) AMPUTATION<br>(PX) | PXCH | 27596 | RE-AMPUTATION OF THIGH THROUGH THIGH BONE | 27596 |
| X_LOWER_AMP | LOWER EXTREMITY<br>(LIMB) AMPUTATION<br>(PX) | PXCH | 27598 | DETACHMENT OF KNEE | 27598 |
| | LOWER EXTREMITY<br>(LIMB) AMPUTATION | | | | |
| X_LOWER_AMP | (PX) | PXCH | 27880 | AMPUTATION OF BOTH LOWER LEG BONES | 27880 |
| PX LOWER AMP | LOWER EXTREMITY<br>(LIMB) AMPUTATION<br>(PX) | PXCH | 27881 | AMPUTATION OF LEG | 27881 |
| 202/\_/\\\ | i , | | 2.001 | 2.7.11011 01 220 | 2.001 |
| PX_LOWER_AMP | LOWER EXTREMITY<br>(LIMB) AMPUTATION<br>(PX) | PXCH | 27882 | AMPUTATION OF LEG, OPEN PROCEDURE | 27882 |
| PX LOWER AMP | LOWER EXTREMITY<br>(LIMB) AMPUTATION<br>(PX) | PXCH | 27884 | AMPUTATION OF LEG, SECONDARY CLOSURE | 27884 |
| | LOWER EXTREMITY (LIMB) AMPUTATION | | | | |
| X LOWER AMP | (PX) | PXCH | 27886 | RE-AMPUTATION OF LEG | 27886 |
| | LOWER EXTREMITY<br>(LIMB) AMPUTATION | | | | |
| PX_LOWER_AMP | (PX) | PXCH | 27888 | AMPUTATION OF FOOT AT ANKLE | 27888 |
| PX LOWER AMP | LOWER EXTREMITY<br>(LIMB) AMPUTATION<br>(PX) | PXCH | 27889 | AMPUTATION OF FOOT THROUGH ANKLE JOINT | 27889 |
| | LOWER EXTREMITY<br>(LIMB) AMPUTATION | | | | |
| PX_LOWER_AMP | (PX) LOWER EXTREMITY (LIMB) AMPUTATION | PXCH | 28800 | AMPUTATION OF MIDFOOT BONE | 28800 |
| PX LOWER AMP | (PX) | PXCH | 28805 | AMPUTATION OF FOOT ACROSS INSTEP | 28805 |
| DY LOWER AMP | LOWER EXTREMITY (LIMB) AMPUTATION (PX) | PXCH | 28810 | AMPLITATION OF TOE AND MIDEOUT PONE | 28810 |
| PX_LOWER_AMP | i , | 1 7011 | 20010 | AMPUTATION OF TOE AND MIDFOOT BONE | 20010 |
| PX_LOWER_AMP | LOWER EXTREMITY<br>(LIMB) AMPUTATION<br>(PX) | PXCH | 28820 | AMPUTATION OF TOE AT JOINT BETWEEN THE FOREFOOT AND TOES | 28820 |
| | LOWER EXTREMITY (LIMB) AMPUTATION | | | | |
| PX_LOWER_AMP | (PX) | PXCH | 28825 | AMPUTATION OF TOE AT TOE JOINTS | 28825 |
| PX_OBS_APNEA | OBSTRUCTIVE SLEEP<br>APNEA (PX) | PXCH | 94660 | INITIATION AND MANAGEMENT OF CONTINUED PRESSURED RESPIRATORY ASSISTANCE BY MASK OR BREATHING TUBE | 94660 |
| PX_OBS_APNEA | OBSTRUCTIVE SLEEP<br>APNEA (PX) | PXCH | A4604 | TUBING WITH INTEGRATED HEATING ELEMENT FOR USE WITH POSITIVE AIRWAY PRESSURE DEVICE | A4604 |
| PX_OBS_APNEA | OBSTRUCTIVE SLEEP<br>APNEA (PX) | PXCH | A7027 | COMBINATION ORAL/NASAL MASK, USED WITH<br>CONTINUOUS POSITIVE AIRWAY PRESSURE<br>DEVICE, EACH | A7027 |
| PX_OBS_APNEA | OBSTRUCTIVE SLEEP<br>APNEA (PX) | PXCH | A7029 | NASAL PILLOWS FOR COMBINATION<br>ORAL/NASAL MASK, REPLACEMENT ONLY, PAIR | A7029 |
| PX OBS APNEA | OBSTRUCTIVE SLEEP<br>APNEA (PX) | PXCH | A7030 | FULL FACE MASK USED WITH POSITIVE AIRWAY PRESSURE DEVICE, EACH | A7030 |


# **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the following state of

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the following state of

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the State o

BI Study Number 1245-0228

c39712001-02

Boehringer Ingelheim

State of the following state of

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the following state of

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim


Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the state o

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

State of the following of the followi

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| PX_PAD | PAD (PX) | PX10 | 04NY4ZZ | RELEASE LOWER ARTERY, PERCUTANEOUS ENDOSCOPIC APPROACH | 04NY4ZZ |
|---|---|---|---|---|---|
| PX PAD | PAD (PX) | PXCH | 35256 | REPAIR OF BLOOD VESSEL OF LEG WITH VEIN GRAFT | 35256 |
| X PAD | PAD (PX) | PXCH | 35286 | REPAIR OF BLOOD VESSEL OF LEG WITH GRAFT | 35286 |
| X PAD | PAD (PX) | PXCH | 35351 | REMOVAL OF BLOOD CLOT AND PORTION OF ARTERY OF GROIN | 35351 |
| _ | | | | REMOVAL OF BLOOD CLOT AND PORTION OF | |
| PX_PAD PX_PAD | PAD (PX) | PXCH | 35355<br>35361 | ARTERY OF UPPER THIGH, ILIOFEMORAL REMOVAL OF BLOOD CLOT AND PORTION OF ARTERY OF ABDOMINAL AORTA AND GROIN ARTERY | 35355<br>35361 |
| X PAD | PAD (PX) | PXCH | 35363 | REMOVAL OF BLOOD CLOT AND PORTION OF<br>ARTERY OF ABDOMINAL AORTA AND UPPER<br>THIGH ARTERY | 35363 |
| X_I/ID<br>PX PAD | PAD (PX) | PXCH | 35371 | REMOVAL OF BLOOD CLOT AND PORTION OF ARTERY OF UPPER THIGH ARTERY, COMMON | 35371 |
| | | | | REMOVAL OF BLOOD CLOT AND PORTION OF | |
| PX_PAD | PAD (PX) | PXCH | 35372 | ARTERY OF UPPER THIGH ARTERY, DEEP | 35372 |
| PX_PAD | PAD (PX) | PXCH | 35381 | THROMBOENDARTERECTOMY, WITH OR WITHOUT PATCH GRAFT; FEMORAL AND/OR POPLITEAL, AND/OR TIBIOPERONEAL | 35381 |
| X_PAD | PAD (PX) | PXCH | 35454 | TRANSLUMINAL BALLOON ANGIOPLASTY, OPEN; ILIAC | 35454 |
| X_PAD | PAD (PX) | PXCH | 35456 | TRANSLUMINAL BALLOON ANGIOPLASTY, OPEN; FEMORAL-POPLITEAL | 35456 |
| X_PAD | PAD (PX) | PXCH | 35459 | TRANSLUMINAL BALLOON ANGIOPLASTY, OPEN;<br>TIBIOPERONEAL TRUNK AND BRANCHES | 35459 |
| PX_PAD | PAD (PX) | PXCH | 35470 | TRANSLUMINAL BALLOON ANGIOPLASTY,<br>PERCUTANEOUS; TIBIOPERONEAL TRUNK OR<br>BRANCHES, EACH VESSEL | 35470 |
| PX_PAD | PAD (PX) | PXCH | 35473 | TRANSLUMINAL BALLOON ANGIOPLASTY, PERCUTANEOUS; ILIAC | 35473 |
| PX_PAD | PAD (PX) | PXCH | 35474 | TRANSLUMINAL BALLOON ANGIOPLASTY, PERCUTANEOUS; FEMORAL-POPLITEAL | 35474 |
| PX_PAD | PAD (PX) | PXCH | 35482 | TRANSLUMINAL PERIPHERAL ATHERECTOMY, OPEN; ILIAC | 35482 |
| PX_PAD | PAD (PX) | PXCH | 35483 | TRANSLUMINAL PERIPHERAL ATHERECTOMY, OPEN; FEMORAL-POPLITEAL | 35483 |
| DV DAD | DAD (DV) | DVOL | 05404 | TRANSLUMINAL PERIPHERAL ATHERECTOMY, OPEN; BRACHIOCEPHALIC TRUNK OR | 05404 |
| PX_PAD | PAD (PX) | PXCH | 35484 | BRANCHES, EACH VESSEL TRANSLUMINAL PERIPHERAL ATHERECTOMY, | 35484 |
| X_PAD | PAD (PX) | PXCH | 35485 | OPEN; TIBIOPERONEAL TRUNK AND BRANCHES TRANSLUMINAL PERIPHERAL ATHERECTOMY, | 35485 |
| PX_PAD | PAD (PX) | PXCH | 35492 | PERCUTANEOUS; ILIAC TRANSLUMINAL PERIPHERAL ATHERECTOMY, | 35492 |
| PX_PAD | PAD (PX) | PXCH | 35493 | PERCUTANEOUS; FEMORAL-POPLITEAL | 35493 |
| PX_PAD | PAD (PX) | PXCH | 35494 | TRANSLUMINAL PERIPHERAL ATHERECTOMY, PERCUTANEOUS; BRACHIOCEPHALIC TRUNK OR BRANCHES, EACH VESSEL | 35494 |
| | . , | | | TRANSLUMINAL PERIPHERAL ATHERECTOMY, PERCUTANEOUS; TIBIOPERONEAL TRUNK AND | |
| PX_PAD | PAD (PX) | PXCH | 35495 | BRANCHES | 35495 |
| X_PAD | PAD (PX) | PXCH | 35521 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(ARM TO UPPER LEG ARTERY), WITH VEIN | 35521 |
| PX_PAD | PAD (PX) | PXCH | 35533 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(ARM TO UPPER LEG AND OPPOSITE LEG<br>ARTERY), WITH VEIN | 35533 |
| PX_PAD | PAD (PX) | PXCH | 35541 | BYPASS GRAFT, WITH VEIN; AORTOILIAC OR<br>BI-ILIAC | 35541 |
| PX PAD | PAD (PX) | PXCH | 35546 | BYPASS GRAFT, WITH VEIN; AORTOFEMORAL OR BIFEMORAL | 35546 |

Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| PX_PAD | PAD (PX) | PXCH | 35548 | BYPASS GRAFT, WITH VEIN;<br>AORTOILIOFEMORAL, UNILATERAL | 35548 |
|---|---|---|---|---|---|
| PX_PAD | PAD (PX) | PXCH | 35549 | BYPASS GRAFT, WITH VEIN;<br>AORTOILIOFEMORAL, BILATERAL | 35549 |
| PX_PAD | PAD (PX) | PXCH | 35551 | BYPASS GRAFT, WITH VEIN;<br>AORTOFEMORAL-POPLITEAL | 35551 |
| PX PAD | PAD (PX) | PXCH | 35556 | BYPASS OF DISEASED OR BLOCKED ARTERY (UPPER TO LOWER LEG ARTERY), WITH VEIN | 35556 |
| PX PAD | PAD (PX) | PXCH | 35558 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(UPPER LEG TO OPPOSITE UPPER LEG ARTERY),<br>WITH VEIN | 35558 |
| PX PAD | PAD (PX) | PXCH | 35560 | BYPASS OF DISEASED OR BLOCKED ARTERY (AORTA TO KIDNEY ARTERY), WITH VEIN | 35560 |
| | | | | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(GROIN TO OPPOSITE GROIN ARTERY), WITH | |
| PX_PAD | PAD (PX) | PXCH | 35563 | VEIN | 35563 |
| PX_PAD | PAD (PX) | PXCH | 35565 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(GROIN TO UPPER LEG ARTERY), WITH VEIN | 35565 |
| PX_PAD | PAD (PX) | PXCH | 35566 | BYPASS OF DISEASED OR BLOCKED ARTERY (UPPER LEG TO LOWER LEG ARTERY), WITH VEIN | 35566 |
| PX PAD | PAD (PX) | PXCH | 35570 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(LOWER LEG TO OPPOSITE LOWER LEG<br>ARTERY), WITH VEIN | 35570 |
| 1 <u>7 1 7 D</u> | I AD (I A) | TACIT | 33370 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(LOWER LEG TO LOWER LEG ARTERY), WITH | 33370 |
| PX_PAD | PAD (PX) | PXCH | 35571 | VEIN | 35571 |
| PX_PAD | PAD (PX) | PXCH | 35582 | | 35582 |
| PX_PAD | PAD (PX) | PXCH | 35583 | BYPASS OF DISEASED OR BLOCKED ARTERY BY INSERTION OF VEIN GRAFT FROM ARTERY OF THIGH TO ARTERY OF KNEE (FEMORAL-POPLITEAL BYPASS) | 35583 |
| PX_PAD | PAD (PX) | PXCH | 35585 | BYPASS OF DISEASED OR BLOCKED ARTERY BY INSERTION OF VEIN GRAFT FROM ARTERY OF THIGH TO ARTERY OF LOWER LEG (FEMORAL-ANTERIOR TIBIAL, POSTERIOR TIBIAL, OR PERONEAL ARTERY BYPASS) | 35585 |
| | | | | BYPASS OF DISEASED OR BLOCKED ARTERY BY<br>INSERTION OF VEIN GRAFT FROM ARTERY OF<br>KNEE TO ARTERY OF LOWER LEG<br>(POPLITEAL-TIBIAL OR PERONEAL ARTERY | |
| PX_PAD | PAD (PX) | PXCH | 35587 | BYPASS) | 35587 |
| PX_PAD | PAD (PX) | PXCH | 35621 | BYPASS OF DISEASED OR BLOCKED ARTERY (ARM TO CHEST ARTERY), OTHER THAN VEIN | 35621 |
| PX PAD | PAD (PX) | PXCH | 35623 | BYPASS OF DISEASED OR BLOCKED ARTERY (ARM TO LOWER LEG ARTERY), OTHER THAN VEIN | 35623 |
| PX_PAD | PAD (PX) | PXCH | 35637 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(AORTA TO GROIN ARTERY), OTHER THAN VEIN | 35637 |
| PX_PAD | PAD (PX) | PXCH | 35638 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(AORTA TO GROIN TO OPPOSITE GROIN<br>ARTERY), OTHER THAN VEIN | 35638 |
| | , , | | | BYPASS GRAFT, WITH OTHER THAN VEIN; | |
| PX_PAD | PAD (PX) | PXCH | 35641 | AORTOILIAC OR BI-ILIAC BYPASS OF DISEASED OR BLOCKED ARTERY | 35641 |
| PX_PAD | PAD (PX) | PXCH | 35646 | (AORTA TO UPPER LEG AND OPPOSITE UPPER<br>LEG ARTERY), OTHER THAN VEIN | 35646 |
| PX_PAD | PAD (PX) | PXCH | 35647 | BYPASS OF DISEASED OR BLOCKED ARTERY (AORTA TO UPPER LEG ARTERY), OTHER THAN VEIN | 35647 |
| PX PAD | PAD (PX) | PXCH | 35650 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(UNDER ARM TO OPPOSITE ARM ARTERY),<br>OTHER THAN VEIN | 35650 |

Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| | | | | BYPASS OF DISEASED OR BLOCKED ARTERY | |
|---|---|---|---|---|---|
| PX_PAD | PAD (PX) | PXCH | 35654 | (ARM TO BOTH LOWER THIGH ARTERIES),<br>OTHER THAN VEIN | 35654 |
| PX_PAD | PAD (PX) | PXCH | 35656 | BYPASS OF DISEASED OR BLOCKED ARTERY (UPPER LEG TO LOWER THIGH ARTERY), OTHER THAN VEIN | 35656 |
| PX_PAD | PAD (PX) | PXCH | 35661 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(UPPER LEG TO OPPOSITE UPPER LEG ARTERY),<br>OTHER THAN VEIN | 35661 |
| PX_PAD | PAD (PX) | PXCH | 35663 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(GROIN TO OPPOSITE GROIN ARTERY), OTHER<br>THAN VEIN | 35663 |
| PX_PAD | PAD (PX) | PXCH | 35665 | BYPASS ON DISEASED OR BLOCKED GROIN TO UPPER LEG ARTERY, OTHER THAN VEIN | 35665 |
| PX_PAD | PAD (PX) | PXCH | 35666 | BYPASS OF DISEASED OR BLOCKED ARTERY<br>(UPPER LEG TO LOWER LEG ARTERIES), OTHER<br>THAN VEIN | 35666 |
| PX_PAD | PAD (PX) | PXCH | 35671 | BYPASS OF DISEASED OR BLOCKED ARTERY (KNEE TO LOWER LEG ARTERIES), OTHER THAN VEIN | 35671 |
| PX_PAD | PAD (PX) | PXCH | 35681 | BYPASS OF DISEASED OR BLOCKED ARTERY, COMPOSITE | 35681 |
| PX_PAD | PAD (PX) | PXCH | 35682 | BYPASS OF DISEASED OR BLOCKED ARTERY, COMPOSITE, 2 VEINS | 35682 |
| PX_PAD | PAD (PX) | PXCH | 35683 | BYPASS OF DISEASED OR BLOCKED ARTERY, COMPOSITE, 3 OR MORE VEINS | 35683 |
| PX_PAD | PAD (PX) | PXCH | 35879 | REVISION OF ARTERIAL BYPASS OF LEG WITH PLACEMENT OF VEIN PATCH, OPEN PROCEDURE | 35879 |
| PX_PAD | PAD (PX) | PXCH | 37207 | INSERTION OF STENT IN BLOOD VESSEL VIA CATHETER | 37207 |
| PX_PAD | PAD (PX) | PXCH | 37208 | INSERTION OF STENT IN BLOOD VESSEL VIA CATHETER | 37208 |
| PX_PAD | PAD (PX) | PXCH | 37220 | BALLOON DILATION OF ARTERY IN ONE SIDE OF<br>GROIN, ENDOVASCULAR, ACCESSED THROUGH<br>THE SKIN OR OPEN PROCEDURE | 37220 |
| PX PAD | PAD (PX) | PXCH | 37221 | INSERTION OF STENTS IN ARTERY IN ONE SIDE OF GROIN, ENDOVASCULAR, ACCESSED THROUGH THE SKIN OR OPEN PROCEDURE | 37221 |
| PX PAD | PAD (PX) | PXCH | 37222 | BALLOON DILATION OF GROIN ARTERY,<br>ENDOVASCULAR, OPEN, OR PERCUTANEOUS<br>APPROACH | 37222 |
| PX PAD | PAD (PX) | PXCH | 37223 | INSERTION OF STENTS INTO GROIN ARTERY,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE | 37223 |
| PX PAD | PAD (PX) | PXCH | 37224 | BALLOON DILATION OF ARTERIES IN ONE LEG,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE | 37224 |
| PX PAD | PAD (PX) | PXCH | 37225 | REMOVAL OF PLAQUE IN ARTERIES IN ONE LEG,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE | 37225 |
| PX PAD | PAD (PX) | PXCH | 37226 | INSERTION OF STENTS INTO ARTERIES IN ONE<br>LEG, ENDOVASCULAR, ACCESSED THROUGH<br>THE SKIN OR OPEN PROCEDURE | 37226 |
| | ( A) | I AGII | 5,220 | REMOVAL OF PLAQUE AND INSERTION OF STENTS INTO ARTERIES IN ONE LEG, | 0,220 |
| PX_PAD | PAD (PX) | PXCH | 37227 | ENDOVASCULAR, ACCESSED THROUGH THE SKIN OR OPEN PROCEDURE | 37227 |
| PX_PAD | PAD (PX) | PXCH | 37228 | BALLOON DILATION OF ARTERY OF ONE LEG,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE | 37228 |
| PX_PAD | PAD (PX) | PXCH | 37229 | REMOVAL OF PLAQUE IN ARTERY IN ONE LEG,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE | 37229 |

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| | | | | INSERTION OF STENTS INTO ARTERY IN ONE<br>LEG, ENDOVASCULAR, ACCESSED THROUGH | |
|---|---|---|---|---|---|
| PX_PAD | PAD (PX) | PXCH | 37230 | THE SKIN OR OPEN PROCEDURE | 37230 |
| PX_PAD | PAD (PX) | PXCH | 37231 | REMOVAL OF PLAQUE AND INSERTION OF<br>STENTS INTO ARTERY IN ONE LEG,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE | 37231 |
| PX_PAD | PAD (PX) | PXCH | 37232 | BALLOON DILATION OF ARTERY IN ONE LEG,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE | 37232 |
| PX PAD | PAD (PX) | PXCH | 37233 | REMOVAL OF PLAQUE IN ARTERY IN ONE LEG,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE, EACH ADDITIONAL<br>VESSEL | 37233 |
| PX_PAD | PAD (PX) | PXCH | 37234 | INSERTION OF STENTS INTO ARTERY IN ONE<br>LEG, ENDOVASCULAR, ACCESSED THROUGH<br>THE SKIN OR OPEN PROCEDURE, EACH<br>ADDITIONAL VESSEL | 37234 |
| PX_PAD | PAD (PX) | РХСН | 37235 | REMOVAL OF PLAQUE AND INSERTION OF<br>STENTS INTO ARTERY IN ONE LEG,<br>ENDOVASCULAR, ACCESSED THROUGH THE<br>SKIN OR OPEN PROCEDURE, EACH ADDITIONAL<br>VESSEL | 37235 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX09 | 00.66 | PERCUTANEOUS TRANSLUMINAL CORONARY<br>ANGIOPLASTY [PTCA] | 66 |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX09 | 17.55 | TRANSLUMINAL CORONARY ATHERECTOMY | 1755 |
| PX PCI | CORONARY REVASCULARIZATION, PCI (PX) | PX09 | 36.01 | TRANSCOMMAN ATTICNED TOWN | 3601 |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX09 | 36.02 | | 3602 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX09 | 36.05 | | 3605 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX09 | 36.06 | INSERTION OF NON-DRUG-ELUTING CORONARY ARTERY STENT(S) | 3606 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX09 | 36.07 | INSERTION OF DRUG-ELUTING CORONARY ARTERY STENT(S) | 3607 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX09 | 36.09 | OTHER REMOVAL OF CORONARY ARTERY OBSTRUCTION | 3609 |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX10 | 0270346 | DILATION OF CORONARY ARTERY, ONE ARTERY,<br>BIFURCATION, WITH DRUG-ELUTING<br>INTRALUMINAL DEVICE, PERCUTANEOUS<br>APPROACH | 270346 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX10 | 027034Z | DILATION OF CORONARY ARTERY, ONE ARTERY WITH DRUG-ELUTING INTRALUMINAL DEVICE, PERCUTANEOUS APPROACH | 027034Z |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX10 | 0270356 | DILATION OF CORONARY ARTERY, ONE ARTERY,<br>BIFURCATION, WITH TWO DRUG-ELUTING<br>INTRALUMINAL DEVICES, PERCUTANEOUS<br>APPROACH | 270356 |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PX10 | 027035Z | DILATION OF CORONARY ARTERY, ONE ARTERY WITH TWO DRUG-ELUTING INTRALUMINAL DEVICES, PERCUTANEOUS APPROACH | 027035Z |

Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| | CORONARY<br>REVASCULARIZATION, | | | BALLOON DILATION OF NARROWED OR<br>BLOCKED MAJOR CORONARY ARTERY OR<br>BRANCH (ACCESSED THROUGH THE SKIN), EACH | |
|---|---|---|---|---|---|
| PX_PCI | PCI (PX) | PXCH | 92920 | ADDITIONAL ARTERY OR BRANCH | 92920 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92921 | BALLOON DILATION OF NARROWED OR BLOCKED MAJOR CORONARY ARTERY OR BRANCH (ACCESSED THROUGH THE SKIN), SINGLE ARTERY OR BRANCH | 92921 |
| DV D01 | CORONARY<br>REVASCULARIZATION, | 2001 | | REMOVAL OF PLAQUE OF MAJOR CORONARY ARTERY OR BRANCH, ACCESSED THROUGH THE | |
| PX_PCI | PCI (PX) | PXCH | 92924 | SKIN, SINGLE ARTERY OR BRANCH | 92924 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92925 | REMOVAL OF PLAQUE OF MAJOR CORONARY<br>ARTERY OR BRANCH, ACCESSED THROUGH THE<br>SKIN, EACH ADDITIONAL ARTERY OR BRANCH | 92925 |
| | CORONARY<br>REVASCULARIZATION, | | | CATHETER PLACEMENT OF STENTS IN MAJOR<br>CORONARY ARTERY OR BRANCH, ACCESSED<br>THROUGH THE SKIN, EACH ADDITIONAL ARTERY | |
| PX_PCI | PCI (PX) | PXCH | 92928 | OR BRANCH | 92928 |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92929 | CATHETER PLACEMENT OF STENTS IN MAJOR<br>CORONARY ARTERY OR BRANCH, ACCESSED<br>THROUGH THE SKIN, SINGLE ARTERY OR<br>BRANCH | 92929 |
| _ | CORONARY<br>REVASCULARIZATION, | | | REMOVAL OF PLAQUE AND INSERTION OF STENT<br>IN MAJOR CORONARY ARTERY OR BRANCH,<br>ACCESSED THROUGH THE SKIN, SINGLE | |
| PX_PCI | PCI (PX) | PXCH | 92933 | ARTERY OR BRANCH | 92933 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92934 | REMOVAL OF PLAQUE AND INSERTION OF STENT<br>IN MAJOR CORONARY ARTIERY OR BRANCH,<br>ACCESSED THROUGH THE SKIN, EACH<br>ADDITIONAL ARTIERY OR BRANCH | 92934 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92937 | INSERTION OF STENT, REMOVAL OF PLAQUE<br>AND/OR BALLOON DILATION OF CORONARY<br>VESSEL, ACCESSED THROUGH THE SKIN,<br>SINGLE VESSEL, INCLUDING DISTAL<br>PROTECTION WHEN PERFORMED | 92937 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92938 | INSERTION OF STENT, REMOVAL OF PLAQUE<br>AND/OR BALLOON DILATION OF CORONARY<br>VESSEL, ACCESSED THROUGH THE SKIN, EACH<br>ADDITIONAL BRANCH | 92938 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92941 | INSERTION OF STENT, REMOVAL OF PLAQUE<br>AND/OR BALLOON DILATION OF CORONARY<br>VESSEL DURING HEART ATTACK, ACCESSED<br>THROUGH THE SKIN | 92941 |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92943 | INSERTION OF STENT, REMOVAL OF PLAQUE<br>AND/OR BALLOON DILATION OF CORONARY<br>VESSEL, ACCESSED THROUGH THE SKIN,<br>SINGLE VESSEL | 92943 |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92944 | INSERTION OF STENT, REMOVAL OF PLAQUE<br>AND/OR BALLOON DILATION OF CORONARY<br>VESSEL, ACCESSED THROUGH THE SKIN, EACH<br>ADDITIONAL ARTERY, BRANCH OR GRAFT | 92944 |
| | CORONARY<br>REVASCULARIZATION, | 1,7,011 | 02011 | TRANSCATHETER PLACEMENT OF AN INTRACORONARY STENT(S), PERCUTANEOUS, WITH OR WITHOUT OTHER THERAPEUTIC | J. 17 |
| PX_PCI | PCI (PX) | PXCH | 92980 | INTERVENTION, ANY METHOD; SINGLE VESSEL TRANSCATHETER PLACEMENT OF AN INTRACORONARY STENT(S), PERCUTANEOUS, WITH OR WITHOUT OTHER THERAPEUTIC | 92980 |
| PX_PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92981 | INTERVENTION, ANY METHOD; EACH<br>ADDITIONAL VESSEL (LIST SEPARATELY IN<br>ADDITION TO CODE FOR PRIMARY PROCEDURE) | 92981 |
| PX PCI | CORONARY<br>REVASCULARIZATION,<br>PCI (PX) | PXCH | 92982 | PERCUTANEOUS TRANSLUMINAL CORONARY<br>BALLOON ANGIOPLASTY; SINGLE VESSEL | 92982 |

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02


DocuSign Envelope ID: 7BE3DD49-FB85-41C7-8861-1DAA3C5DD479

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02

| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 50630 | REMOVAL OF STONE FROM LOWER URINARY DUCT (URETER) | 50630 |
|---|---|---|---|---|---|
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 50945 | REMOVAL OF STONE FROM URINARY DUCT (URETER) USING AN ENDOSCOPE | 50945 |
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 50961 | REMOVAL OF FOREIGN BODY OR STONE FROM KIDNEY OR URINARY DUCT (URETER) USING AN ENDOSCOPY WHICH IS INSERTED THROUGH AN ALREADY CREATED URINARY DUCT (URETER) OPENING | 50961 |
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 50980 | REMOVAL OF FOREIGN BODY OR STONE FROM KIDNEY OR URINARY DUCT (URETER) USING AN ENDOSCOPE | 50980 |
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 51060 | INCISION OF BLADDER WITH REMOVAL OF STONE IN URINARY DUCT (URETER) | 51060 |
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 51065 | INCISION OF BLADDER WITH BASKET REMOVAL<br>AND/OR ULTRASONIC CRUSHING OF STONES IN<br>URINARY DUCT (URETER) | 51065 |
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 52320 | REMOVAL OF STONE IN URINARY DUCT (URETER) USING AN ENDOSCOPE | 52320 |
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 52325 | FRAGMENTING OF STONE IN URINARY DUCT (URETER) USING AN ENDOSCOPE | 52325 |
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 52352 | REMOVAL OR MANIPULATION OF STONE IN URINARY DUCT (URETER) OR KIDNEY USING AN ENDOSCOPE | 52352 |
| PX_STONE_KID | KIDNEY STONE (PX) | PXCH | 52353 | CRUSHING OF STONE IN URINARY DUCT (URETER) USING AN ENDOSCOPE | 52353 |

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study (NIS)

BI Study Number 1245-0228

c39712001-02


Boehringer Ingelheim

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study
(NIS)

BI Study Number 1245-0228

c39712001-02


#### **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| CONCEPT_ID | CONCEPT_LBL | DRUG_INPUT |
|-----------------------------|-----------------------------|------------------|
| MD_ACE | ACE INHIBITORS | BENAZEPRIL |
| MD_ACE | ACE INHIBITORS | CAPTOPRIL |
| MD_ACE | ACE INHIBITORS | ENALAPRIL |
| MD_ACE | ACE INHIBITORS | FOSINOPRIL |
| MD_ACE | ACE INHIBITORS | LISINOPRIL |
| MD ACE | ACE INHIBITORS | MOEXIPRIL |
| MD ACE | ACE INHIBITORS | PERINDOPRIL |
| MD ACE | ACE INHIBITORS | QUINAPRIL |
| MD ACE | ACE INHIBITORS | RAMIPRIL |
| MD ACE | ACE INHIBITORS | TRANDOLAPRIL |
| MD AGI | ALPHA-GLUCOSIDASE INHIBITOR | ACARBOSE |
| MD AGI | ALPHA-GLUCOSIDASE INHIBITOR | MIGLITOL |
| MD ALPHA BLOCK | ALPHA BLOCKERS | DOXAZOSIN |
| MD ALPHA BLOCK | ALPHA BLOCKERS | PRAZOSIN |
| MD_ALPHA_BLOCK | ALPHA BLOCKERS | TERAZOSIN |
| MD_ALITIA_BLOCK MD_AMYLINO | AMYLINOMIMETIC | PRAMLINTIDE |
| _ | | |
| MD_ANTICONV | ANTICONVULSANTS | ALPRAZOLAM |
| MD_ANTICONV | ANTICONVULSANTS | BRIVARACETAM |
| MD_ANTICONV | ANTICONVULSANTS | CANNABIDIOL |
| MD_ANTICONV | ANTICONVULSANTS | CARBAMAZEPINE |
| MD_ANTICONV | ANTICONVULSANTS | CENOBAMATE |
| MD_ANTICONV | ANTICONVULSANTS | CHLORDIAZEPOXIDE |
| MD_ANTICONV | ANTICONVULSANTS | CLONAZEPAM |
| MD_ANTICONV | ANTICONVULSANTS | CLORAZEPATE |
| MD_ANTICONV | ANTICONVULSANTS | DIAZEPAM |
| MD_ANTICONV | ANTICONVULSANTS | ESLICARBAZEPINE |
| MD_ANTICONV | ANTICONVULSANTS | ETHOSUXIMIDE |
| MD_ANTICONV | ANTICONVULSANTS | FELBAMATE |
| MD_ANTICONV | ANTICONVULSANTS | FOSPHENYTOIN |
| MD_ANTICONV | ANTICONVULSANTS | GABAPENTIN |
| MD_ANTICONV | ANTICONVULSANTS | LACOSAMIDE |
| MD_ANTICONV | ANTICONVULSANTS | LAMOTRIGINE |
| MD_ANTICONV | ANTICONVULSANTS | LEVETIRACETAM |
| MD_ANTICONV | ANTICONVULSANTS | LORAZEPAM |
| MD_ANTICONV | ANTICONVULSANTS | OXAZEPAM |
| MD_ANTICONV | ANTICONVULSANTS | OXCARBAZEPINE |
| MD ANTICONV | ANTICONVULSANTS | PERAMPANEL |
| MD ANTICONV | ANTICONVULSANTS | PHENOBARBITAL |
| MD ANTICONV | ANTICONVULSANTS | PHENYTOIN |
| MD ANTICONV | ANTICONVULSANTS | PREGABALIN |
| MD ANTICONV | ANTICONVULSANTS | PRIMIDONE |
| MD ANTICONV | ANTICONVULSANTS | RUFINAMIDE |
| MD ANTICONV | ANTICONVULSANTS | STIRIPENTOL |
| MD_ANTICONV | ANTICONVULSANTS | TIAGABINE |
| MD ANTICONV | ANTICONVULSANTS | TOPIRAMATE |
| MD_ANTICONV | ANTICONVULSANTS | VALPROATE |
| MD_ANTICONV | ANTICONVULSANTS | |
| _ | | VIGABATRIN |
| MD_ANTICONV | ANTICONVULSANTS | ZONISAMIDE |
| MD_ANTIDEP | ANTIDEPRESSANTS | AMOVADINE |
| MD_ANTIDEP | ANTIDEPRESSANTS | AMOXAPINE |
| MD_ANTIDEP | ANTIDEPRESSANTS | BUPROPION |
| MD_ANTIDEP | ANTIDEPRESSANTS | CITALOPRAM |
| MD_ANTIDEP | ANTIDEPRESSANTS | DESIPRAMINE |
| MD_ANTIDEP | ANTIDEPRESSANTS | DESVENLAFAXINE |
| MD ANTIDEP | ANTIDEPRESSANTS | DOXEPIN |


#### **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| MD_ANTIDEP | ANTIDEPRESSANTS | DULOXETINE |
|--------------------------------|---------------------|-----------------|
| MD ANTIDEP | ANTIDEPRESSANTS | ESCITALOPRAM |
| MD ANTIDEP | ANTIDEPRESSANTS | FLUOXETINE |
| MD ANTIDEP | ANTIDEPRESSANTS | FLUVOXAMINE |
| MD ANTIDEP | ANTIDEPRESSANTS | ISOCARBOXAZID |
| MD ANTIDEP | ANTIDEPRESSANTS | LEVOMILNACIPRAN |
| MD ANTIDEP | ANTIDEPRESSANTS | MAPROTILINE |
| MD ANTIDEP | ANTIDEPRESSANTS | MIRTAZAPINE |
| MD ANTIDEP | ANTIDEPRESSANTS | NEFAZODONE |
| MD ANTIDEP | ANTIDEPRESSANTS | NORTRIPTYLINE |
| MD_ANTIDEP | ANTIDEPRESSANTS | PAROXETINE |
| MD ANTIDEP | ANTIDEPRESSANTS | PHENELZINE |
| MD ANTIDEP | ANTIDEPRESSANTS | PROTRIPTYLINE |
| MD ANTIDEP | ANTIDEPRESSANTS | SERTRALINE |
| MD_ANTIDEP | ANTIDEPRESSANTS | TRANYLCYPROMINE |
| MD_ANTIDEP | ANTIDEPRESSANTS | TRAZODONE |
| MD_ANTIDEP | ANTIDEPRESSANTS | VENLAFAXINE |
| MD_ANTIDEP | ANTIDEPRESSANTS | VILAZODONE |
| MD_ANTIDEP | ANTIDEPRESSANTS | VORTIOXETINE |
| | ANTIPLATELET AGENTS | ABCIXIMAB |
| MD_ANTIP | | ASPIRIN |
| MD_ANTIP | ANTIPLATELET ACENTS | |
| MD_ANTIP | ANTIPLATELET AGENTS | CANGRELOR |
| MD_ANTIP | ANTIPLATELET ACENTS | CLOPIDOGREL |
| MD_ANTIP | ANTIPLATELET AGENTS | EPTIFIBATIDE |
| MD_ANTIP | ANTIPLATELET AGENTS | PRASUGREL |
| MD_ANTIP | ANTIPLATELET AGENTS | TICAGRELOR |
| MD_ANTIP | ANTIPLATELET AGENTS | TIROFIBAN |
| MD_ANTIP | ANTIPLATELET AGENTS | VORAPAXAR |
| MD_ANTIPSY | ANTIPSYCHOTICS | ARIPIPRAZOLE |
| MD_ANTIPSY | ANTIPSYCHOTICS | ASENAPINE |
| MD_ANTIPSY | ANTIPSYCHOTICS | BREXPIPRAZOLE |
| MD_ANTIPSY | ANTIPSYCHOTICS | CARIPRAZINE |
| MD_ANTIPSY | ANTIPSYCHOTICS | CHLORPROMAZINE |
| MD_ANTIPSY | ANTIPSYCHOTICS | CLOZAPINE |
| MD_ANTIPSY | ANTIPSYCHOTICS | FLUPHENAZINE |
| MD_ANTIPSY | ANTIPSYCHOTICS | HALOPERIDOL |
| MD_ANTIPSY | ANTIPSYCHOTICS | ILOPERIDONE |
| MD_ANTIPSY | ANTIPSYCHOTICS | LOXAPINE |
| MD_ANTIPSY | ANTIPSYCHOTICS | LUMATEPERONE |
| MD_ANTIPSY | ANTIPSYCHOTICS | LURASIDONE |
| MD_ANTIPSY | ANTIPSYCHOTICS | OLANZAPINE |
| MD_ANTIPSY | ANTIPSYCHOTICS | PALIPERIDONE |
| MD ANTIPSY | ANTIPSYCHOTICS | PERPHENAZINE |
| MD ANTIPSY | ANTIPSYCHOTICS | QUETIAPINE |
| MD ANTIPSY | ANTIPSYCHOTICS | RISPERIDONE |
| MD ANTIPSY | ANTIPSYCHOTICS | THIORIDAZINE |
| MD_ANTIPSY | ANTIPSYCHOTICS | THIOTHIXENE |
| MD ANTIPSY | ANTIPSYCHOTICS | TRIFLUOPERAZINE |
| MD ANTIPSY | ANTIPSYCHOTICS | ZIPRASIDONE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | ACEBUTOLOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | ADENOSINE |
| MD_ANTI_ARRYTH | ANTIARRHYTHMICS | AMIODARONE |
| MD_ANTI_ARRYTH | ANTIARRHYTHMICS | ATENOLOL |
| MD_ANTI_ARRYTH | ANTIARRHYTHMICS | BETAXOLOL |
| MD_ANTI_ARRYTH MD_ANTI_ARRYTH | ANTIARRHYTHMICS | BISOPROLOL |
| MP VIXII VI/L/1111 | ANTAKKITITIMIOO | BISOFROLOL |


## **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| MD_ANTI_ARRYTH | ANTIARRHYTHMICS | DIGOXIN |
|---|---|---|
| MD_ANTI_ARRYTH | ANTIARRHYTHMICS | DILTIAZEM |
| MD_ANTI_ARRYTH | ANTIARRHYTHMICS | DISOPYRAMIDE |
| MD_ANTI_ARRYTH | ANTIARRHYTHMICS | DOFETILIDE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | DRONEDARONE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | ESMOLOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | FLECAINIDE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | IBUTILIDE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | LABETALOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | LIDOCAINE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | METOPROLOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | MEXILETINE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | NADOLOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | NEBIVOLOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | PINDOLOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | PROCAINAMIDE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | PROPAFENONE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | PROPRANOLOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | QUINIDINE |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | SOTALOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | TIMOLOL |
| MD ANTI ARRYTH | ANTIARRHYTHMICS | VERAPAMIL |
| MD ARB | ANGIOTENSIN II RECEPTOR BLOCKERS | AZILSARTAN |
| MD ARB | ANGIOTENSIN II RECEPTOR BLOCKERS | CANDESARTAN |
| MD ARB | ANGIOTENSIN II RECEPTOR BLOCKERS | EPROSARTAN |
| MD ARB | ANGIOTENSIN II RECEPTOR BLOCKERS | IRBESARTAN |
| MD ARB | ANGIOTENSIN II RECEPTOR BLOCKERS | LOSARTAN |
| MD ARB | ANGIOTENSIN II RECEPTOR BLOCKERS | OLMESARTAN |
| MD ARB | ANGIOTENSIN II RECEPTOR BLOCKERS | TELMISARTAN |
| MD_ARB | ANGIOTENSIN II RECEPTOR BLOCKERS | VALSARTAN |
| MD_ARB | ARNI | SACUBITRIL |
| MD ASTHMA COPD | COPD OR ASTHMA MEDICATIONS | ACLIDINIUM |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | ALBUTEROL |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | ARFORMOTEROL<br>RECLOMETHAS ONE |
| MD_ASTHMA_COPD | COPD OR ASTUMA MEDICATIONS | BECLOMETHASONE |
| MD_ASTHMA_COPD | COPD OR ASTUMA MEDICATIONS | BENRALIZUMAB |
| MD_ASTHMA_COPD | COPD OR ASTUMA MEDICATIONS | BUDESONIDE |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | CICLESONIDE |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | DUPILUMAB |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | FLUTICASONE |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | FORMOTEROL |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | GLYCOPYRRONIUM |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | INDACATEROL |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | IPRATROPIUM |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | LEVALBUTEROL |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | MEPOLIZUMAB |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | MOMETASONE |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | MONTELUKAST |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | OLODATEROL |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | OMALIZUMAB |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | RESLIZUMAB |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | REVEFENACIN |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | ROFLUMILAST |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | SALMETEROL |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | THEOPHYLLINE |
| MD ASTHMA COPD | COPD OR ASTHMA MEDICATIONS | TIOTROPIUM |


## **Boehringer Ingelheim** Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | UMECLIDINIUM |
|---|---|---|
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | VILANTEROL |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | ZAFIRLUKAST |
| MD_ASTHMA_COPD | COPD OR ASTHMA MEDICATIONS | ZILEUTON |
| MD BB | BETA BLOCKERS | ACEBUTOLOL |
| MD BB | BETA BLOCKERS | ATENOLOL |
| MD BB | BETA BLOCKERS | BETAXOLOL |
| MD BB | BETA BLOCKERS | BISOPROLOL |
| MD BB | BETA BLOCKERS | CARVEDILOL |
| MD BB | BETA BLOCKERS | ESMOLOL |
| MD BB | BETA BLOCKERS | LABETALOL |
| MD BB | BETA BLOCKERS | METOPROLOL |
| MD BB | BETA BLOCKERS | NADOLOL |
| MD BB | BETA BLOCKERS | NEBIVOLOL |
| MD_BB | BETA BLOCKERS | PINDOLOL |
| MD_BB | BETA BLOCKERS | PROPRANOLOL |
| MD BB | | |
| | BETA BLOCKERS | TIMOLOL |
| MD_BENZOD | BENZODIAZEPINES | ALPRAZOLAM |
| MD_BENZOD | BENZODIAZEDINES | CHLORDIAZEPOXIDE |
| MD_BENZOD | BENZODIAZEPINES | CLONAZEPAM |
| MD_BENZOD | BENZODIAZEPINES | CLORAZEPATE |
| MD_BENZOD | BENZODIAZEPINES | DIAZEPAM |
| MD_BENZOD | BENZODIAZEPINES | LORAZEPAM |
| MD_BENZOD | BENZODIAZEPINES | OXAZEPAM |
| MD_BISPHO | BISPHOSPHONATES | ALENDRONATE |
| MD_BISPHO | BISPHOSPHONATES | IBANDRONATE |
| MD_BISPHO | BISPHOSPHONATES | RISEDRONATE |
| MD_BISPHO | BISPHOSPHONATES | ZOLEDRONIC |
| MD_CCB | CALCIUM CHANNEL BLOCKERS | AMLODIPINE |
| MD_CCB | CALCIUM CHANNEL BLOCKERS | CLEVIDIPINE |
| MD_CCB | CALCIUM CHANNEL BLOCKERS | FELODIPINE |
| MD CCB | CALCIUM CHANNEL BLOCKERS | ISRADIPINE |
| MD CCB | CALCIUM CHANNEL BLOCKERS | NICARDIPINE |
| MD CCB | CALCIUM CHANNEL BLOCKERS | NIFEDIPINE |
| MD CCB | CALCIUM CHANNEL BLOCKERS | NIMODIPINE |
| MD CCB | CALCIUM CHANNEL BLOCKERS | NISOLDIPINE |
| MD_CCB_ND | CALCIUM CHANNEL BLOCKERS - NON-DIHYDROPYRIDINE | DILTIAZEM |
| MD CCB ND | CALCIUM CHANNEL BLOCKERS - NON-DIHYDROPYRIDINE | VERAPAMIL |
| MD CIPR | CIPROFLOXACIN | CIPROFLOXACIN |
| MD DEMENTIA | DEMENTIA MEDICATIONS | DONEPEZIL |
| MD DEMENTIA | DEMENTIA MEDICATIONS | GALANTAMINE |
| MD DEMENTIA | DEMENTIA MEDICATIONS | MEMANTINE |
| MD DEMENTIA | DEMENTIA MEDICATIONS | RIVASTIGMINE |
| | | DIGOXIN |
| MD_DIGOXIN | DIGOXIN | |
| MD_DPP4 | DIPERTIDYL PERTIDASE 4 (DPP4) INHIBITOR | ALOGLIPTIN |
| MD_DPP4 | DIPEPTIDYL PEPTIDASE-4 (DPP4) INHIBITOR | LINAGLIPTIN |
| MD_DPP4 | DIPEPTIDYL PEPTIDASE-4 (DPP4) INHIBITOR | SAXAGLIPTIN |
| MD_DPP4 | DIPEPTIDYL PEPTIDASE-4 (DPP4) INHIBITOR | SITAGLIPTIN |
| MD_EMPA | EMPAGLIFLOZIN | EMPAGLIFLOZIN |
| MD_FINEREN | FINERENONE | FINERENONE |
| MD_FLUCO | FLUCONAZOLE | FLUCONAZOLE |
| MD_GLITAZONE | GLITAZONE | PIOGLITAZONE |
| MD_GLITAZONE | GLITAZONE | ROSIGLITAZONE |
| MD_GLP1 | GLUCAGON-LIKE PEPTIDE-1 (GLP1) RECEPTOR AGONIST | ALBIGLUTIDE |
| MD_GLP1 | GLUCAGON-LIKE PEPTIDE-1 (GLP1) RECEPTOR AGONIST | DULAGLUTIDE |
| MD_GLP1 | GLUCAGON-LIKE PEPTIDE-1 (GLP1) RECEPTOR AGONIST | EXENATIDE |

Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| MD GLP1 | GLUCAGON-LIKE PEPTIDE-1 (GLP1) RECEPTOR AGONIST | LIRAGLUTIDE |
|---|---|---|
| MD GLP1 | GLUCAGON-LIKE PEPTIDE-1 (GLP1) RECEPTOR AGONIST | LIXISENATIDE |
| MD_GLF1 | GLUCAGON-LIKE PEPTIDE-1 (GLP1) RECEPTOR AGONIST | SEMAGLUTIDE |
| MD HEPARIN | HEPARIN AND OTHER LMWH | DALTEPARIN |
| MD HEPARIN | HEPARIN AND OTHER LIMWH | ENOXAPARIN |
| _ | HEPARIN AND OTHER LIMWH | |
| MD_HEPARIN | | HEPARIN |
| MD_INSULIN | INSULIN | ASPART |
| MD_INSULIN | INSULIN | DEGLUDEC |
| MD_INSULIN | INSULIN | DETEMIR |
| MD_INSULIN | INSULIN | GLARE |
| MD_INSULIN | INSULIN | GLARGINE |
| MD_INSULIN | INSULIN | GLULISINE |
| MD_INSULIN | INSULIN | LISPRO |
| MD_INSULIN | INSULIN | NPH |
| MD_INSULIN | INSULIN | REGULAR |
| MD_LEVO | LEVOFLOXACIN | LEVOFLOXACIN |
| MD_LOOP | LOOP DIURETICS | BUMETANIDE |
| MD_LOOP | LOOP DIURETICS | ETHACRYNATE |
| MD_LOOP | LOOP DIURETICS | FUROSEMIDE |
| MD_LOOP | LOOP DIURETICS | TORSEMIDE |
| MD_MEGLI | MEGLINITIDES | NATEGLINIDE |
| MD_MEGLI | MEGLINITIDES | REPAGLINIDE |
| MD_METFORMIN | METFORMIN | METFORMIN |
| MD_MOXI | MOXIFLOXACIN | MOXIFLOXACIN |
| MD NITR | NITROFURANTOIN | NITROFURANTOIN |
| MD NITRATE | NITRATES | ISOSORBIDE |
| MD NITRATE | NITRATES | NITROGLYCERIN |
| MD NORF | NORFLOXACIN | NORFLOXACIN |
| MD NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | ASPIRIN |
| MD NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | CELECOXIB |
| MD NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | DICLOFENAC |
| MD NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | ETODOLAC |
| MD NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | IBUPROFEN |
| MD NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | INDOMETHACIN |
| MD NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | KETOROLAC |
| MD NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | MELOXICAM |
| MD NSAID | | NABUMETONE |
| | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | |
| MD_NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | NAPROXEN |
| MD_NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | PIROXICAM |
| MD_NSAID | NONSTEROIDAL ANTI-INFLAMMATORY DRUGS | SULINDAC |
| MD_OPIOIDS | OPIOIDS | CODEINE |
| MD_OPIOIDS | OPIOIDS | FENTANYL |
| MD_OPIOIDS | OPIOIDS | HYDROCODONE |
| MD_OPIOIDS | OPIOIDS | HYDROMORPHONE |
| MD_OPIOIDS | OPIOIDS | MEPERIDINE |
| MD_OPIOIDS | OPIOIDS | METHADONE |
| MD_OPIOIDS | OPIOIDS | MORPHINE |
| MD_OPIOIDS | OPIOIDS | OXYCODONE |
| MD_OPIOIDS | OPIOIDS | OXYMORPHONE |
| MD_ORALCORT | ORAL CORTICOSTEROIDS | BETAMETHASONE |
| MD_ORALCORT | ORAL CORTICOSTEROIDS | CORTISONE |
| MD_ORALCORT | ORAL CORTICOSTEROIDS | DEXAMETHASONE |
| MD_ORALCORT | ORAL CORTICOSTEROIDS | HYDROCORTISONE |
| MD ORALCORT | ORAL CORTICOSTEROIDS | METHYLPREDNISOLONE |
| MD_ORALCORT | ORAL CORTICOSTEROIDS | PREDNISOLONE |
| MD ORALCORT | ORAL CORTICOSTEROIDS | PREDNISONE |

Boehringer Ingelheim  Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| MD_ORALCORT | ORAL CORTICOSTEROIDS | TRIAMCINOLONE |
|---|---|---|
| MD_ORAL_COAG | ORAL ANTICOAGULANTS | APIXABAN |
| MD_ORAL_COAG | ORAL ANTICOAGULANTS | BETRIXABAN |
| MD_ORAL_COAG | ORAL ANTICOAGULANTS | DABIGATRAN |
| MD ORAL COAG | ORAL ANTICOAGULANTS | EDOXABAN |
| MD ORAL COAG | ORAL ANTICOAGULANTS | RIVAROXABAN |
| MD ORAL COAG | ORAL ANTICOAGULANTS | WARFARIN |
| MD OTHER DIURETIC | OTHER DIURETICS | AMILORIDE |
| MD OTHER DIURETIC | OTHER DIURETICS | EPLERENONE |
| MD OTHER DIURETIC | OTHER DIURETICS | SPIRONOLACTONE |
| MD OTHER DIURETIC | OTHER DIURETICS | TRIAMTERENE |
| MD OTHER HTN | OTHER HYPERTENSION DRUGS | ALISKIREN |
| MD OTHER HTN | OTHER HYPERTENSION DRUGS | CLONIDINE |
| MD_OTHER_HTN | OTHER HYPERTENSION DRUGS | HYDRALAZINE |
| MD OTHER HTN | OTHER HYPERTENSION DRUGS | METHYLDOPA |
| MD_OTHER_HTN | OTHER HYPERTENSION DRUGS | MINOXIDIL |
| MD OTHER LIPID | OTHER LIPID LOWERING DRUGS | ALIROCUMAB |
| MD OTHER LIPID | OTHER LIPID LOWERING DRUGS | CHOLESTYRAMINE |
| MD_OTHER_LIPID | OTHER LIPID LOWERING DRUGS | COLESEVELAM |
| MD OTHER LIPID | OTHER LIPID LOWERING DRUGS | COLESTIPOL |
| MD OTHER LIPID | OTHER LIPID LOWERING DRUGS | EVOLOCUMAB |
| MD OTHER LIPID | OTHER LIPID LOWERING DRUGS | EZETIMIBE |
| MD OTHER LIPID | OTHER LIPID LOWERING DRUGS | FENOFIBRATE |
| MD_OTHER_LIPID | OTHER LIPID LOWERING DRUGS | GEMFIBROZIL |
| MD_OTHER_LIPID | OTHER LIPID LOWERING DRUGS | NIACIN |
| MD OT ANX HYP | OTHER ANXIOLYTICS OR HYPNOTICS | AMOBARBITAL |
| | OTHER ANXIOLYTICS OR HYPNOTICS OTHER ANXIOLYTICS OR HYPNOTICS | BUSPIRONE |
| MD_OT_ANX_HYP | | |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | ESZOPICLONE |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | FLURAZEPAM |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | METHOHEXITAL |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | PENTOBARBITAL |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | QUAZEPAM |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | RAMELTEON |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | SECOBARBITAL |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | TEMAZEPAM |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | THIOPENTAL |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | TRIAZOLAM |
| MD_OT_ANX_HYP | OTHER ANXIOLYTICS OR HYPNOTICS | ZOLPIDEM |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | ABATACEPT |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | ADALIMUMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | ANAKINRA |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | AZATHIOPRINE |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | BASILIXIMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | CERTOLIZUMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | CYCLOSPORINE |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | DACLIZUMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | ETANERCEPT |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | EVEROLIMUS |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | GOLIMUMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | INFLIXIMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | IXEKIZUMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | LEFLUNOMIDE |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | MYCOPHENOLATE |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | NATALIZUMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | RITUXIMAB |
| MD OT IMMSUP | OTHER IMMUNOSUPPRESSIVES | SECUKINUMAB |

Boehringer Ingelheim 
Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Study

BI Study Number 1245-0228

c39712001-02

| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | SIROLIMUS |
|---|---|---|
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | TACROLIMUS |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | TOCILIZUMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | TOFACITINIB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | USTEKINUMAB |
| MD_OT_IMMSUP | OTHER IMMUNOSUPPRESSIVES | VEDOLIZUMAB |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | AMANTADINE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | APOMORPHINE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | BENZTROPINE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | CARBIDOPA |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | DROXIDOPA |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | ENTACAPONE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | ISTRADEFYLLINE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | PRAMIPEXOLE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | RASAGILINE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | ROPINIROLE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | ROTIGOTINE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | SAFINAMIDE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | SELEGILINE |
| MD_PARKINSON | ANTIPARKINSONIAN MEDICATIONS | TRIHEXYPHENIDYL |
| MD_SGLT2 | SODIUM-GLUCOSE TRANSPORT PROTEIN 2 (SGLT2) INHIBITOR | CANAGLIFLOZIN |
| MD_SGLT2 | SODIUM-GLUCOSE TRANSPORT PROTEIN 2 (SGLT2) INHIBITOR | DAPAGLIFLOZIN |
| MD_SGLT2 | SODIUM-GLUCOSE TRANSPORT PROTEIN 2 (SGLT2) INHIBITOR | ERTUGLIFLOZIN |
| MD_STATIN | STATINS | ATORVASTATIN |
| MD_STATIN | STATINS | FLUVASTATIN |
| MD_STATIN | STATINS | LOVASTATIN |
| MD_STATIN | STATINS | PITAVASTATIN |
| MD_STATIN | STATINS | PRAVASTATIN |
| MD_STATIN | STATINS | ROSUVASTATIN |
| MD_STATIN | STATINS | SIMVASTATIN |
| MD_SULF | SULFAMETHOXAZOLE | SULFAMETHOXAZOLE |
| MD_SULFONYLUREA | SULFONYLUREA | GLIMEPIRIDE |
| MD_SULFONYLUREA | SULFONYLUREA | GLIPIZIDE |
| MD_SULFONYLUREA | SULFONYLUREA | GLYBURIDE |
| MD_THIAZIDE | THIAZIDE DIURETICS | CHLOROTHIAZIDE |
| MD_THIAZIDE | THIAZIDE DIURETICS | CHLORTHALIDONE |
| MD_THIAZIDE | THIAZIDE DIURETICS | INDAPAMIDE |
| MD_THIAZIDE | THIAZIDE DIURETICS | METOLAZONE |



#### APPROVAL / SIGNATURE PAGE

Document Number: c39712001 Technical Version Number: 2.0

**Document Name:** 8-01-seap

**Title:** Comparative cardiovascular and renal effectiveness and safety of Empagliflozin and other SGLT2i in patients with type 2 diabetes (T2D), with and without baseline kidney disease in the United States

# **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|--------------------------------|-----------|------------------------|
| Approval-Clinical Trial Leader | | 02 Aug 2023 15:11 CEST |
| Approval | | 14 Aug 2023 19:25 CEST |

Boehringer IngelheimPage 2 of 2Document Number: c39712001Technical Version Number:2.0

(Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | <b>Date Signed</b> |
|----------------------|-----------|--------------------|
|----------------------|-----------|--------------------|